## **Document Coversheet**

Study Title: Transcranial Magnetic Stimulation (TMS) for Smoking Cessation in People Living With HIV/AIDS (PLWHA)

| Institution/Site: | University of Kentucky |
|----------------------------------|---------------------------------|
| Document (Approval/Update) Date: | 2/7/2023 (IRB); 2/24/2022 (ICF) |
| NCT Number: | NCT04936594 |
| IRB Number | 64473 |
| Coversheet created: | 4/4/2023 |

### **PROTOCOL TYPE (VERSION 4)**

IRB Approval 2/7/2023
IRB # 64473
IRB3
CLOSED

| -Which IRB- |
|------------------------------------------------|
| െ Medical േ NonMedical |
| Protocol Process Type |
| • • |
| © Exemption © Expedited (Must be risk level 1) |
| Full |
| G I UII |

IMPORTANT NOTE: You will not be able to change your selections for "Which IRB" and "Protocol Process Type" after saving this section. If you select the wrong IRB or Protocol Process Type, you may need to create a new application.

See below for guidance on these options, or refer to ORI's "Getting Started" page. Please contact the Office of Research Integrity (ORI) at 859-257-9428 with any questions prior to saving your selections.

#### \*Which IRB\*

The Medical IRB reviews research from the Colleges of:

- Dentistry
- · Health Sciences
- Medicine
- Nursing
- Pharmacy and Health Sciences
- and Public Health.

The Nonmedical IRB reviews research from the Colleges of:

- Agriculture
- · Arts and Sciences
- · Business and Economics
- Communication and Information
- · Design; Education
- · Fine Arts
- Law
- and Social Work

**Note:** Studies that involve administration of drugs, testing safety or effectiveness of medical devices, or invasive medical procedures must be reviewed by the **Medical IRB** regardless of the college from which the application originates.

#### \*Which Protocol Process Type\*

Under federal regulations, the IRB can process an application to conduct research involving human subjects in one of three ways:

- by exemption certification
- · by expedited review.
- · by full review;

The investigator makes the preliminary determination of the type of review for which a study is eligible. Please refer to ORI's "Getting Started" page for more information about which activities are eligible for each type of review.

The revised Common Rule expanded exemption certification category 4 for certain secondary research with identifiable information or biospecimens. The regulations no longer require the information or biospecimens to be existing. For more information see the <u>Exemption Categories Tool</u>.

#### **CONTINUATION REVIEW/FINAL REVIEW**

0 unresolved comment(s)

Based on your responses to the Continuation Review/Final Review questions, to be in accord with federal policy a final review report must be submitted to properly CLOSE OUT your protocol. IF YOU WISH TO EXTEND YOUR IRB APPROVAL PERIOD, update your 'Anticipated Ending Date of Research Project' under the Project Information section and include any other supportive documentation for continuation of your study [NOTE: If you wish for your IRB approval to continue, but you do not request an extension and complete and submit your materials in a timely manner, IRB approval will expire at the end of the current approval period.].

If you have any questions, please contact the Office of Research Integrity at 859-257-9428.



To initiate your continuation review (CR)/annual administrative review (AAR), or properly close your study, complete this section and update/correct all other sections of your IRB application as applicable.

\*\*\*IMPORTANT\*\*\* Before leaving this page to update other sections of your application, be sure to SAVE this section first.

#### 1. Status of the Research

Check the statement(s) that best describe(s) the current status of your research: •

- □ No subjects have enrolled to date.
- □ Recruitment and/or enrollment of new subjects or review of records/specimens continue.
- □ Study is closed to enrollment, but subjects still receive research-related interventions (e.g., treatment, blood draws).
- □ Study enrollment is permanently closed; subjects have completed all research-related interventions; and the study remains active only for long-term follow-up of subjects (see Tool Tip above for info on long-term follow-up of subjects).\*
- □ Research has progressed to the point that it involves 1) Data analysis, including analysis of identifiable private information or identifiable biospecimens; and/or 2) Accessing follow-up clinical data from procedures that subjects would undergo as part of clinical care.\*
- □The remaining research activities are limited only to data analysis. There is access to records or specimens either directly or through codes or links to the data.\*
- □The remaining research activities are limited only to data analysis. There is no subject/record/specimen identifying codes or links to the data; the researcher or research team cannot readily ascertain the subject's identity.\*
- \*Possibility that review will move from Full to Expedited.
- 2. If subjects have been enrolled within the last year, and the IRB approved a consent/assent form for your study, attach one copy of the entire signed consent/assent form/HIPAA form for the last TWO subjects enrolled.



#### 3. Informed Consent

If the study is open to subject enrollment, please go to the Informed Consent section of the E-IRB Application and verify attachment(s) include:

- One clean copy in PDF (without the IRB Approval stamp) of the currently approved consent/assent document(s), or,
- If requesting changes to the consent/assent document(s), submit one copy with the changes highlighted (and designate Document Type as "Highlighted"), and one clean copy in PDF (without the changes highlighted).

If the study is open to subject enrollment and the IRB has waived the requirement to document informed consent, please go to the Informed Consent section of the E-IRB Application and verify attachment(s) include:

- One clean copy in PDF of the currently approved document used for the informed consent process (e.g., cover letter, phone script), or,
- If requesting changes to the consent/assent document(s), submit one copy with the changes highlighted (and designate Document Type as "Highlighted"), and one clean copy in PDF (without the changes highlighted).

If the study is closed to subject enrollment, please go to the Informed Consent section of the E-IRB Application and remove Informed Consent Documents designated to get an IRB approval stamp to avoid having them appear valid for enrollment.

### 4. Unanticipated Problems Involving Risk to Subjects or Others/Adverse Events Summary & Assessment

| c Yes ⊚ No |
|---|
| n the space below, provide a written summary of both unanticipated problems* and available information regarding adverse events |
| since the last review (e.g., initial review or annual/continuing review). The amount of detail provided in such a summary will vary |

in the space below, provide a written summary of both unanticipated problems" and available information regarding adverse events since the last review (e.g., initial review or annual/continuing review). The amount of detail provided in such a summary will vary depending on the type of research being conducted; in many cases, such a summary could be a brief statement that there have been no unanticipated problems and that adverse events have occurred at the expected frequency and level of severity as documented in the research protocol, the informed consent document, and investigator's brochure (if applicable). The summary must include the Pl's assessment whether the problems/adverse events warrant changes to the protocol, consent process, or risk/benefit ratio.

Note: It is the IRB's expectation that all unanticipated problems involving risk to subjects or others or related deaths requiring prompt reporting are submitted in the appropriate time frame (See Policy [PDF]). Your response to this Annual/Continuing Review is considered assurance that all prompt reportable problems/adverse events have been submitted for IRB review.

| 5. Subject Info To-Date |
|---|
| Our records for the previously approved IRB application indicate the <b>IRB approved estimate</b> of subjects to be enrolled (or records/specimens reviewed) is: |
| 60 |
| Enter the number of enrolled subjects (or records/specimens reviewed) that have not been previously reported to the IRB |
| 0 |
| Our records for the previously approved IRB application indicate the previous total # of subjects enrolled (or records/specimens reviewed) since activation of the study is: 9 |
| The new total number of subjects enrolled (or records/specimens reviewed) since activation of the study: 9 |
| Please review the Project Info section for the IRB approved estimate of subjects to be enrolled (or records/specimens reviewed). If this new total exceeds your approved estimate of subjects to be enrolled (or records/specimens reviewed), please update the number in the field for Number of Human Subjects in the Project Info section. |

### 6. Data and Safety Monitoring Board (DSMB)/Plan (DSMP)

Did any problems/adverse events occur during the last 12 months?

If your study is monitored by a DSMB or under a DSMP, attach all documentation (i.e. summary report; meeting minutes) representing Data and Safety Monitoring activities that have not been previously reported to the IRB.

Attachments

#### 7. Since the most recent IRB Initial/Continuation Review Approval:

Have there been any **participant complaints** regarding the research?

C Yes © No

If yes, in the field below, provide a summary describing the complaints.

Have any **subjects withdrawn** from the research voluntarily or by you as the PI for reasons related to safety, welfare, or problems related to the conduct of the research? If a participant does not meet the screening criteria for a study even if they signed a screening

<sup>\*</sup>For multisite studies, the written summary should describe external events determined to be unanticipated problems involving risk to subjects or others.

consent it is NOT considered a withdrawal.

∩ Yes ∩ No

If yes, in the field below, provide a detailed explanation to the withdrawal(s) including if participants were lost to contact.

Has any **new and relevant literature** been published since the last IRB review, especially literature relating to risks associated with the research?

Yes 
 No

If yes, attach a copy of the literature as well as a brief summary of the literature including, if pertinent, the impact of the findings on the protection of human subjects.

#### Attachments

Have there been any interim findings?

Yes No

If yes, attach a copy of Interim Findings.

#### Attachments

#### Have subjects experienced any benefits?

∩ Yes ∈ No

If yes, in the field below, provide a description of benefits subjects have experienced.

Have there been any **inspections/audits/quality improvement reviews** of your research protocol resulting in the need for corrective action in order to protect the safety and welfare of subjects?

∩ Yes @ No

If yes, please attach documentation evidencing the outcome(s) and any corrective action(s) taken as a result.

### Attachments

Was an FDA 483 issued as a result of any inspections/audits?

If yes, submit documentation using attachment button above.

### 8. Risk Level:

Our records for the previously approved IRB application show your research is:

Risk Level: 2

Has something during the course of your research changed the level of risk?

∩ Yes @ No

If yes, go to the Risk Level section, mark the appropriate risk level, and in the field below, describe why the risk level has changed:

### 9. Funding/Support:

Our records for the **previously approved I**RB application indicate your research is being submitted to, supported by, or conducted in cooperation with the following external or internal agency(ies) or funding program(s):

■ Grant application pending

■ (HHS) Dept. of Health & Human Services

**(NIH)** National Institutes of Health

□ (CDC) Centers for Disease Control & Prevention

| | 64473 |
|---|---|
| ☐ (HRSA) Health Resources and Services Administration | CLOSED |
| □ (SAMHSA) Substance Abuse and Mental Health Services Administration | |
| □ (DoJ) Department of Justice or Bureau of Prisons | |
| □ (DoE) Department of Energy | |
| □ (EPA) Environmental Protection Agency | |
| ■ Federal Agencies Other Than Those Listed Here | |
| □ Industry (Other than Pharmaceutical Companies) | |
| ✓ Internal Grant Program w/ proposal | |
| □ Internal Grant Program w/o proposal | |
| ☐ National Science Foundation | |
| □ Other Institutions of Higher Education | |
| □ Pharmaceutical Company | |
| ☐ Private Foundation/Association | |
| □ U.S. Department of Education | |
| <b>□</b> State | |
| Other | |

Please **update the Funding/Support section of your IRB application** if needed, including the following attachments if they contain changes not previously reported to the IRB:

- A current copy of your protocol if you are conducting industry/pharmaceutical research;
- A current Investigator Brochure (submit a copy with all changes underlined).
- A new or revised grant application for this project.

Did your project receive extramural funding?

⊂ Yes ∈ No

If yes, please review and correct if necessary, the OSPA Account # information under the **Funding/Support section** of your IRB application.

If the project is externally funded, has the sponsor offered any of the research team enrollment incentives or other personal benefit bonuses? (e.g., cash/check, travel reimbursements, gift checks, etc.)

∩ Yes ∩ No ⊚ N/A

Note: It is University of Kentucky policy that personal benefit bonuses are not allowed. If these conditions change during the course of the study, please notify the IRB.

#### 10. Project Information

Our records for the previously approved IRB application indicate your estimated project end date is:

### 03/30/2024

If you have a new estimated project end date, please go to the Project Info section and change the date in the field for Anticipated Ending Date of Research Project.

### 11. Study Personnel

Our records for the previously approved IRB application indicate the following individuals are study personnel on this project (if applicable):

| Last Name | First Name |
|-----------|------------|
| Thornton | Alice |
| Christian | Amy |
| Rush | Craig |
| Jasinski | Lindsey |
| Burris | Jessica |
| Su | Amanda |

| Last Name | First Name |
|--------------------|------------|
| Bell | Robert |
| Garth | Patricia |
| Cordero | Patrick |
| Anand | Pavan |
| Wesley | Michael |
| Kahl | Joan |
| Alcorn | Joseph |
| Khanal | Rebika |
| Elias | Madona |
| Hime <b>l</b> hoch | Seth |
| Adams Jr. | Thomas |
| Sabitus | Kathryn |

Please review the individuals listed above and update your records as needed in the Study Personnel section of the E-IRB application, being sure that each individual listed has completed or is up-to-date on the mandatory human research protection training [see the policy on <u>Mandatory Human Subject Protection Training FAQs</u> (required every three years)].

### 12. Progress of the Research

To meet federal requirements the IRB is relying on your RESEARCH DESCRIPTION as a protocol summary and their expectation is that it is up-to-date. If the currently approved protocol (or research description) in your E-IRB application is outdated, please make applicable changes, and describe in the field below any substantive changes and explain why they are essential. If none, insert "N/A" in the text field below. If you are closing your study, you may use the space below to summarize the final status of the research.

We enrolled nine participants. With the preliminary findings, we could submit an extramural grant application to the National Institute of Drug Abuse (NIDA). Therefore, we will would like to close this IRB.

Thank you,

Gopalkumar, Rakesh, MD

Note: No changes in the research procedures should have occurred without previous IRB review. Approval from the IRB must be obtained before implementing any changes.

Provide a brief summary of any modifications that affect subject safety and/or welfare approved by the IRB since the last initial or continuation review (If none, insert "N/A" in the text field below.):

N/A

Attach one copy of the most recent progress report sent to the FDA, if available. All PI-sponsored IND/IDE studies are required to submit a copy of the FDA progress report.

Attachments

#### 13. Confidentiality/Security

Review your Research Description section and update the Confidentiality portion, if necessary, to describe measures for security of electronic and physical research records (e.g., informed consent document(s), HIPAA Authorization forms, sensitive or private data).

### 14. Subject Demographics

# Our records for the previously approved IRB application indicate the following categories of subjects a included in your research:

- Children (individuals under age 18)
- **■** Wards of the State (Children)
- **■** Emancipated Minors
- Students
- **■** College of Medicine Students
- **UK Medical Center Residents or**

House Officers

- Impaired Consent Capacity Adults
- Pregnant Women/Neonates/Fetal

Material

- Prisoners
- Non-English Speaking
- International Citizens
- Normal Volunteers
- Military Personnel and/or DoD

Civilian Employees

- **■** Patients
- Appalachian Population

Please review the Subject Demographics section of your IRB application for accuracy, and note the following:

If during the course of your research 1) any prisoners have been enrolled, OR 2) subjects have been enrolled that became involuntarily confined/detained in a penal institution that have not been previously reported to the IRB, go to Subject Demographic section in your E-IRB application and mark "prisoners" in the categories of subjects to be included in the study, if it is not already marked.

Note: If either 1 or 2 above apply, and you have received funding from the Department of Health and Human Services (HHS), a Certification Letter should have been submitted to the Office for Human Research Protections (OHRP); prisoners and individuals who have become involuntarily confined/detained in a penal institution cannot continue participation in the research until OHRP issues approval. If the Certification has not been submitted, contact the Office of Research Integrity.

Based on the total # of subjects who have enrolled, complete the subject demographic section below:

| Participant Demographics | | | | |
|---|---|---|---|---|
| | Cisgender Man 🕕 | Cisgender Woman 🕡 | TGNB/TGE 🕡 | Unknown/Not Reported |
| American | | | | |
| idian/A <b>l</b> askan | | | | |
| Native <sup>-</sup> | | | | |
| Asian | | | | |
| Black or | | | | |
| African | 2 | | | |
| American | | | | |
| Latinx | | | | |
| Native | | | | |
| Hawaiian or | | | | |
| Other Pacific | | | | |
| Islander | | | | |
| White | 1 | 1 | | |
| American | | | | |
| Arab/Middle | | | | |
| Eastern/North | | | | |
| African | | | | |
| Indigenous | | | | |
| People | | | | |
| Around the Wor <b>l</b> d | | | | |
| More than | | 1 | | |
| One Race | | | | |

| lf unknown, please explain why: | |
|---|---|
| 5. Research Sites | |
| Our records for the previously approved IRB application indicate that | t you are conducting research at the following sites: |
| UK Sites | 1 |
| □ UK Classroom(s)/Lab(s) | |
| ■ UK Clinics outside of Lexington | |
| ☐ UK Healthcare Good Samaritan Hospital | |
| □ UK Hospital | |
| Schools/Education Institutions Schools/Education | |
| Institutions | |
| ■ Fayette Co. School Systems * | |
| ☐ Other State/Regional School Systems | |
| ■Institutions of Higher Education (other than UK) | |
| | ] |

Other Medical Facilities

Unknown or Not Reported

- Bluegrass Regional Mental Health Retardation Board
- □ Cardinal Hill Hospital
- Eastern State Hospital
- Nursing Homes
- Shriner's Children's Hospital
- Other Hospitals and Med. Centers
- Correctional Facilities
- Home Health Agencies
- International Sites

Other:

If the above listed sites are not accurate, go to the Research Sites section of the E-IRB application to update the facilities at which research procedures have been or will be conducted.

If you are adding a new off-site facility, you may also need to update your E-IRB application Research Description, Research Sites, Informed Consent, and other affected sections as well as any documents which will list the off-site facility. Documents needing updating may include, but not limited to:

- Consent forms (attachment under Informed Consent section)
- Brochures (attachment under Additional Info section)
- Advertisements (attachment under Research Description section);
- Letter of support (attachment under Research Sites section)).

Please revise applicable sections and attachments as necessary.

### 16. Disclosure of Significant Financial Interest

Disclosure of Significant Financial Interest:

Our records for the previously approved IRB application indicate that you, your investigators, and/or key personnel (KP) have a significant financial interest (SFI) related to your/their responsibilities at the University of Kentucky (that requires disclosure per the UK administrative regulation 7:2):

If you need to update your records, please go to the PI Contact Information section and/or Details for individuals listed in the Study Personnel section to change your response to the applicable question(s).

### 17. Supplementals

To ensure the IRB has the most accurate information for your protocol you are expected to re-visit the E-IRB application sections and make corrections or updates as needed. At a minimum you are being asked to review the following sections for accuracy:

STUDY DRUG INFORMATION—Please review for accuracy. STUDY DEVICE INFORMATION—Please review for accuracy. RESEARCH ATTRIBUTES—Please review for accuracy. OTHER REVIEW COMMITTEES -- Please review for accuracy.

If applicable, submit one copy of the entire signed HIPAA Authorization form for the same last TWO subjects enrolled.

Attachments

### PROJECT INFORMATION

0 unresolved comment(s)

| Title of Project: (Use the exact title listed in the grant/contract application, if applicable). If your research investigates any aspect of COVID-19, please include "COVID19" at the beginning of your Project Title and Short Title •• |
|---|
| Transcranial Magentic Stimulation (TMS) for Smoking Cessation in People Living with HIV/AIDS (PLWHA) |
| Short Title Description Please use a few key words to easily identify your study - this text will be displayed in the Dashboard listing for your study. |
| TMS for Smoking Cessation in PLWHA |
| Anticipated Ending Date of Research Project: 3/30/2024 |
| Maximum number of human subjects (or records/specimens to be reviewed) 60 |
| After approval, will the study be open to enrollment of new subjects or new data/specimen collection? |

#### PI CONTACT INFORMATION

0 unresolved comment(s)

#### Principal Investigator (PI) role for E-IRB access

The PI is the individual holding primary responsibility on the research project with the following permissions on the E-IRB application:

- Read
- 2. write/edit;
- 3. receive communications; and
- 4. submit to the IRB (IR, CR, MR, Other Review\*).

If research is being submitted to or supported by an extramural funding agency such as NIH, a private foundation or a pharmaceutical/manufacturing company, the PI listed on the grant application or the drug protocol must be listed as PI here.

Please fill in any blank fields with the appropriate contact information (gray shaded fields are not editable). Required fields left blank will be highlighted in pink after you click "Save".

To change home and work addresses, go to <u>myUK</u> and update using the Employee Self Service (ESS) portal. If name has changed, the individual with the name change will need to submit a <u>'Name Change Form'</u> to the Human Resources Benefits Office for entering into SAP. The new name will need to be associated with the individual's Link Blue ID in SAP before the change is reflected in E-IRB. Contact the <u>HR Benefits Office</u> for additional information.

The Principal Investigator's (PI) contact information is filled in automatically based on who logged in to create the application.

#### If you are not the Principal Investigator, do NOT add yourself as study personnel.

To change the PI contact information on an application in Researcher edit status:

- click "Change Principal Investigator";
- search for the PI's name using the search feature;
- click "Select" by the name of the Principal Investigator, then "Save Contact Information".

You will automatically be added as study personnel with editing permissions to continue editing the application.



#### **Change Principal Investigator:**

| E: 1N | | | |
|---|---|---|---|
| First Name: | Gopalkumar | Room# &<br>Bldg: Fount | ain Court |
| Last Name: | Rakesh | Speed<br>Sort#: 1 40509 | 9 |
| Middle Name | | | |
| Department: | Psychiatry - 7H800 | Dept Code: 7H80 | 0 |
| Pľs | | Rank: 🕕 | |
| Employee/Student<br>ID#: | 12461687 | | Assistant Professor |
| Pl's Telephone #: | 857-222-2276 | Degree: | MD |
| PI's e-mail<br>address: | Gopalkumar.Rakesh@uky.edu | PI's FAX<br>Number: | |
| PI is R.N. | ⊂Yes ∘ No | HSP Trained: | Yes |
| | | HSP Trained<br>Date: | 9/15/2022 |
| | | RCR Trained: | Yes |
| | a <u>significant financial interest</u> related<br>K administrative regulation 7:2)? | to your responsibilities at the U | Iniversity of Kentucky (that requires |

0 unresolved comment(s)

-Indicate which of the categories listed below accurately describes this protocol-

- (Risk Level 1) Not greater than minimal risk
- ে (Risk Level 2) Greater than minimal risk, but presenting the prospect of direct benefit to individual subjects
- c (Risk Level 3) Greater than minimal risk, no prospect of direct benefit to individual subjects, but likely to yield generalizable knowledge about the subject's disorder or condition.
- c (Risk Level 4) Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of subjects.
- \*"Minimal risk" means that the probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves from those ordinarily encountered in daily life or during the performance of routine physical or psychological examination or tests.

Refer to <u>UK's quidance document</u> on assessing the research risk for additional information.



**RISK LEVEL** 

0 unresolved comment(s)

#### SUBJECT DEMOGRAPHICS

Age level of human subjects: (i.e., 6 mths.; 2yrs., etc..) 18 to 55

#### Study Population:

Describe the characteristics of the subject population, including age range, gender, ethnic background and health status. Identify the criteria for inclusion and exclusion.

Provide the following information:

- A description of the subject selection criteria and rationale for selection in terms of the scientific objectives and proposed study design;
- A compelling rationale for proposed exclusion of any sex/gender or racial/ethnic group;
- Justification for the inclusion of vulnerable groups such as children, prisoners, adults with impaired consent capacity, or others who may be vulnerable to coercion or undue influence.

Please consider these resources:

NIH Diversity Policy

FDA Diversity Guidance

### Pilot study

Inclusion criteria. Potential participants will be heathy controls who are employed in and around 245 Fountain Court. For inclusion in the pilot, they need to be 1) 18-55 years of age; 2) male or female gender 3) Able to read, understand and communicate in English; 4) Can have a past/current history of smoking. Exclusion criteria. Intoxication with substances on day of the study.

#### Study Proper

Inclusion criteria. Potential participants will be: 1) Patients enrolled in the Bluegrass Clinic; 2) 18-55 years of age; 3) male or female gender 4) Able to read, understand and communicate in English; 5) willing to adhere to the general rules of the Bluegrass Clinic/SMARTClinic/Beyond Birth Clinic; 6) willing and able to abstain from drug use other than Suboxone; 7) exhaled breath on day of study CO < 5 ppm; 8) Stabilized on maintenance buprenoprphine if having comorbid opioid use disorder.

Exclusion criteria. Traumatic brain injury, history of seizure disorder, history of or current diagnosis of schizophrenia, intracranial metal shrapnel, previous adverse effect with TMS, sub-threshold consistency while performing behavioral tasks, failure to show baseline attentional bias to smoking versus neutral cues.

We will exclude pregnant females in our study due to danger of MRI radiation to the unborn fetus.

The main study is not connected to the Bluegrass HIV clinic, SMART clinic or the Beyond Birth Clinic. A person can be enrolled and receiving care at these clinics, and their participation in the research project does not impact their standing in any of these clinics. Participation is truly voluntary in nature.

#### Attachments

Indicate the targeted/planned enrollment of the following members of minority groups and their subpopulations. Possible demographic sources: <u>Census Regional Analyst Edition, Kentucky Race/Ethnic Table, Kentucky Population Data</u>.

(Please note: The IRB will expect this information to be reported at Continuation Review time for Pre-2019 FDA-regulated Expedited review and Full review applications):

| Participant Demographics | | | | |
|---|---|---|---|---|
| | Cisgender Man 📵 | Cisgender Woman 📵 | TGNB/TGE 📵 | Unknown/Not Reported |
| American | | | | |
| Indian/Alaskan<br>Native: | | | | |
| Asian: | | | | |
| Black/African | 2 | | | |
| American: | 3 | | | |
| Latinx: | | | | |
| Native | | | | |
| Hawaiian/Pacific<br>Islander: | | | | |
| | 5 | | | |
| White: | 5 | 1 | | |
| American<br>Arab/Middle | | | | |
| Eastern/North | | | | |
| African: | | | | |
| Indigenous<br>People Around | | | | |
| the World: | | | | |
| More than One | | | | |
| Race: | | | | |
| Unknown or Not Reported: | | | | |

If unknown, please explain why:

Indicate the categories of subjects and controls to be included in the study. You may be required to complete additional forms depending on the subject categories which apply to your research. If the study does not involve direct intervention or direct interaction with subjects, (e.g., record-review research, outcomes registries), do not check populations which the research does not specifically target. For example: a large record review of a diverse population may incidentally include a prisoner or an international citizen, but you should not check those categories if the focus of the study has nothing to do with that status.

Check All That Apply (at least one item must be selected)

#### ADDITIONAL INFORMATION:

- ☐ Children (individuals under age 18)
- ☐ Wards of the State (Children)
- □ Emancipated Minors
- □ Students
- □ College of Medicine Students
- ☐ UK Medical Center Residents or House Officers
- □Impaired Consent Capacity Adults
- ☐ Pregnant Women/Neonates/Fetal Material
- □ Prisoners
- ☐ Non-English Speaking (translated long or short form)
- □ International Citizens
- □ Normal Volunteers
- ☐ Military Personnel and/or DoD Civilian Employees
- Patients
- □ Appalachian Population

- Please visit the <u>IRB Survival Handbook</u> for more information on:
  - Children/Emancipated Minors
  - Students as Subjects
  - Prisoners
  - Impaired Consent Capacity Adults
  - Economically or Educationally Disadvantaged Persons

#### Other Resources:

- UKMC Residents or House Officers [see requirement of GME]
- Non-English Speaking [see also the E-IRB Research Description section on this same topic]
- <u>International Citizens</u> [<u>DoD SOP</u> may apply]
- Military Personnel and/or DoD Civilian Employees

#### Assessment of the potential recruitment of subjects with impaired consent capacity (or likelihood):

Check this box if your study does NOT involve direct intervention or direct interaction with subjects (e.g., record-review research, secondary data analysis). If there is no direct intervention/interaction you will not need to answer the impaired consent capacity questions.

Does this study focus on adult subjects with any conditions that present a high *likelihood* of impaired consent capacity or *fluctuations* in consent capacity? (see examples below)

Yes ○ No

If Yes and you are not filing for exemption certification, go to "Form T", complete the form, and attach it using the button below.

#### Examples of such conditions include:

- Traumatic brain injury or acquired brain injury
- Severe depressive disorders or Bipolar disorders
- Schizophrenia or other mental disorders that
- involve serious cognitive disturbances
- Stroke
- Developmental disabilities
- Degenerative dementias
- CNS cancers and other cancers with possible CNS involvement
- Late stage Parkinson's Disease

- Late stage persistent substance dependence
- Ischemic heart disease
- HIV/AIDS
- COPD
- · Renal insufficiency
- Diabetes
- Autoimmune or inflammatory disorders
- Chronic non-malignant pain disorders
- Drug effects
- Other acute medical crises

#### Attachments

Attach Type File Name
ImpairedConsent Form\_T\_3Ai.doc

#### INFORMED CONSENT/ASSENT PROCESS/WAIVER

0 unresolved comment(s)

For creating your informed consent attachment(s), please download the most up-to-date version listed in "All Templates" under the APPLICATION LINKS menu on the left, and edit to match your research project.

#### Additional Resources:

- Informed Consent/Assent Website
- Waiver of Consent vs. Waiver of Signatures
- Sample Repository/Registry/Bank Consent Template

#### Consent/Assent Tips:

- If you have multiple consent documents, be sure to upload each individually (not all in a combined file).
- If another site is serving as the IRB for the project, attach the form as a "Reliance Consent Form" so the document will not receive a UK IRB approval stamp; the reviewing IRB will need to stamp the consent forms.
- Changes to consent documents (e.g., informed consent form, assent form, cover letter, etc...) should be reflected in a 'tracked changes' version and uploaded separately with the Document Type "Highlighted Changes".
- It is very important that only the documents you wish to have approved by the IRB are attached; DELETE OUTDATED FILES previously approved versions will still be available in Protocol History.
- Attachments that are assigned a Document Type to which an IRB approval stamp applies will be considered the version(s) to be used for enrolling subjects once IRB approval has been issued.
   Document Types that do NOT get an IRB approval stamp are:
  - · "Highlighted Changes",
  - · "Phone Script", and
  - "Reliance Consent Form",
  - "Sponsor's Sample Consent Form".

#### How to Get the Section Check Mark

- 1. You must:
  - a) provide a response in the text box below describing how investigators will obtain consent/assent, and
  - b) check the box for at least one of the consent items and/or check mark one of the waivers
- 2. If applicable attach each corresponding document(s) as a PDF.
- 3. If you no longer need a consent document approved (e.g., closed to enrollment), or, the consent document submitted does not need a stamp for enrolling subjects (e.g., umbrella study, or sub-study), only select "Stamped Consent Doc(s) Not Needed".
- 4. After making your selection(s) be sure to scroll to the bottom of this section and SAVE your work!



### Check All That Apply-

- ▼ Informed Consent Form (and/or Parental Permission Form and/or translated short form)
- ☐ Assent Form
- ☐ Cover Letter (for survey/questionnaire research)
- □ Phone Script
- □ Informed Consent/HIPAA Combined Form
- □ Debriefing and/or Permission to Use Data Form
- □ Reliance Consent Form
- □ Sponsor's sample consent form for Dept. of Health and Human Services (DHHS)-approved protocol
- ☐ Stamped Consent Doc(s) Not Needed

#### Attachments

| Attach Type | File Name |
|---|---|
| Informed Consent/HIPAA Combined Form | Consent_form_Pilot_study_clean copy_V2.pdf |
| Informed Consent/Parental Permission | 64473_Consent_form_TMS_Smoking_V4_clean.pdf |
| Phone Script | 64473_phone_script.pdf |

#### **Informed Consent Process:**

Using active voice, describe how investigators will obtain consent/assent. Include:

- the circumstances under which consent will be sought and obtained
- the timing of the consent process (including any waiting period between providing information and obtaining consent)
- · who will seek consent
- how you will minimize the possibility of coercion or undue influence
- the method used for documenting consent
- if applicable, who is authorized to provide permission or consent on behalf of the subject
- if applicable, specific instruments or techniques to assess and confirm potential subjects' understanding of the information

Note: all individuals authorized to obtain informed consent should be designated as such in the E-IRB "Study Personnel" section of this application.

Special considerations may include:

- · Obtaining consent/assent for special populations such as children, prisoners, or people with impaired decisional capacity
- Research Involving Emancipated Individuals

If you plan to enroll some or all prospective subjects as emancipated, consult with UK legal counsel **prior to submitting this application to the IRB**. Include research legal counsel's recommendations in the "Additional Information" section as a separate document.

- Research Involving Non-English Speaking Subjects
   For information on inclusion of non-English speaking subjects, or subjects from a foreign culture, see IRB Application Instructions for Recruiting Non-English Speaking Participants or Participants from a Foreign Culture.
- Research Repositories

If the purpose of this submission is to establish a research repository describe the informed consent process. For guidance regarding consent issues, process approaches, and sample language see the <u>Sample Repository/Registry/Bank Consent Template</u>.

Informed consent will be obtained after thorough discussion of the research project for both the pilot study and the study proper, what is required of the participant, the risks and benefits of participation in the study, and the procedures that are in place if/when challenges arise. This will be done by the PI, one of the co-investigators or research assistant during the first encounter with the subject, if they fulfill all eligibility criteria and are interested in study participation.

The research project is not connected to the Bluegrass HIV clinic/SMART clinic or Beyond Birth clinic. A person can be enrolled in these clinics and their participation in the research project does not impact their standing in the SMART clinic and therefore the participation is truly voluntary in nature.

If you have questions about the study, you can contact the principal investigator for the study Gopalkumar Rakesh at 857-222-2276. If you have concerns or questions about your rights and/or welfare as a volunteer in this research, you can contact the staff in the Office of Research Integrity at The University of Kentucky at (859) 257-9428 or toll free at 1-866-400-9428. We will give you a signed copy of this consent form to take with you

#### □ Request for Waiver of Informed Consent Process

If you are requesting IRB approval to waive the requirement for the informed consent process, or to alter some or all of the elements of informed consent, complete, Section 1 and Section 2 below.

Note: The IRB does not approve waiver or alteration of the consent process for greater than minimal risk research, except for planned emergency/acute care research as provided under FDA regulations. Contact ORI for regulations that apply to single emergency use waiver or acute care research waiver (859-257-9428).

#### **SECTION 1.**

Check the appropriate item:

■I am requesting a waiver of the requirement for the informed consent process.

■I am requesting an alteration of the informed consent process.

If you checked the box for this item, describe which elements of consent will be altered and/or omitted, and justify the alteration.

#### **SECTION 2.**

Explain how each condition applies to your research.

- a) The research involves no more than minimal risk to the subject.
- b) The rights and welfare of subjects will not be adversely affected.
- c) The research could not practicably be carried out without the requested waiver or alteration.

d) Whenever possible, the subjects or legally authorized representatives will be provided with additional pertiral after they have participated in the study.

- e) If the research involves using or accessing identifiable private information or identifiable biospecimens, the research could not practicably be carried out without using such information or biospecimens in an identifiable format.
  - Private information/specimens are "identifiable" if the investigator may ascertain the identity of the subject or if identifiers
    are associated with the information (e.g., medical records). This could be any of the <u>18 HIPAA identifiers</u> including <u>dates</u>
    of service.
  - If not using identifiable private information or identifiable biospecimens, insert N/A below.

If you are requesting IRB approval to waive the requirement for signatures on informed consent forms, your research activities must fit into one of three regulatory options:

- 1. The only record linking the participant and the research would be the consent document, and the principal risk would be potential harm resulting from a breach of confidentiality (e.g., a study that involves participants who use illegal drugs).
- 2. The research presents no more than minimal risk to the participant and involves no procedures for which written consent is normally required outside of the research context (e.g., a cover letter on a survey, or a phone script).
- 3. The participant (or legally authorized representative) is a member of a distinct cultural group or community in which signing forms is not the norm, the research presents no more than minimal risk to the subject, and there is an appropriate alternative mechanism for documenting that informed consent was obtained.

Select the option below that best fits your study.

If the IRB approves a waiver of signatures, participants must still be provided oral or written information about the study. To ensure you include required elements in your consent document, use the **Cover Letter Template** as a guide. There is an <u>English</u> and a <u>Spanish</u> version.



### Option 1

#### Describe how your study meets these criteria:

- a) The only record linking the participant and the research would be the consent document:
- b) The principal risk would be potential harm resulting from a breach of confidentiality (i.e., a study that involves subjects who use illegal drugs).

Under this option, each participant (or legally authorized representative) must be asked whether (s)he wants to sign a consent document; if the participant agrees to sign a consent document, only an IRB approved version should be used.

#### Option 2

#### Describe how your study meets these criteria:

- a) The research presents no more than minimal risk to the participant:
- b) Involves no procedures for which written consent is normally required outside of the research context (i.e. a cover letter on a survey, or a phone script):

#### Option 3

#### Describe how your study meets these criteria:

- a) The subject (or legally authorized representative) is a member of a distinct cultural group or community in which signing forms is not the norm.
- b) The research presents no more than minimal risk to the subject.
- c) There is an appropriate alternative mechanism for documenting that informed consent was obtained.

STUDY PERSONNEL 0 unresolved comment(s)

Do you have study personnel who will be assisting with the research?

After selecting 'Yes' or 'No' you must click the 'Save Study Personnel Information' button.

Yes a No

-Manage Study Personnel-

Identify other study personnel assisting in research project:

- The individual listed as PI in the 'PI Contact Information' section should NOT be added to this section.
- If the research is required for a University of Kentucky academic program, the faculty advisor is also considered study personnel and should be listed below.

  \*\*\*Residents and students who are PI's are encouraged to designate the faculty advisor or at least one other individual as a contact with an editor role (DP).

  \*\*\*Residents and students who are PI's are encouraged to designate the faculty advisor or at least one other individual as a contact with an editor role (DP).
- Role: DP = Editor (individual can view, navigate, and edit the application for any review phase (IR, CR/FR, MR) or 'Other Review", and submit Other Reviews on behalf of the PI.)
- Role: SP = Reader (individual can view and navigate through the currently approved application only.)

To add an individual via the below feature:

- · Search for personnel;
- Click "select" by the listing for the person you want to add;
- For each person, specify responsibility in the project, whether authorized to obtain informed consent, AND denote who should receive E-IRB notifications (contact status).

NOTE: Study personnel must complete human subject protection (HSP) and Responsible Conduct of Research (RCR) training before implementing any research procedures. For information about training requirements for study personnel, visit UK's HSP FAQ page, the RCR Getting Started page, or contact ORI at 859-257-9428. If you have documentation of current HSP training other than that acquired through UK CITI, you may submit it to ORI (HSPTrainingSupport@uky.edu) for credit.

#### Study personnel assisting in research project: 0

| Last<br>Name | First<br>Name | Responsibility In<br>Project | Role | A<br>C | Contact | Degree | StatusFlag | (HSP) | (HSP)Date | (RCR) | Removed? | Last<br>Updated | SFI |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Adams Jr. | Thomas | Co-Investigator | SP | Υ | N | | Р | Υ | 08/18/2022 | Υ | N | 02/05/2021 | N |
| Alcorn | Joseph | Co-Investigator | DP | Υ | N | PhD | Р | Υ | 05/14/2020 | Υ | N | 02/05/2021 | N |
| Anand | Pavan | Data<br>Analysis/Processing | SP | Υ | N | MD | Р | Υ | 10/18/2022 | Υ | N | 12/28/2022 | N |
| Bell | Robert | Recruitment | SP | Ν | N | | Р | Υ | 01/31/2022 | Υ | N | 07/10/2021 | N |
| Cordero | Patrick | Data<br>Analysis/Processing | SP | Υ | N | MD | Р | Υ | 11/02/2022 | Υ | N | 12/28/2022 | N |
| Elias | Madona | Data<br>Analysis/Processing | DP | N | N | MSW | Р | Υ | 07/18/2022 | Υ | N | 12/28/2022 | N |
| Garth | Patricia | Study Coordinator | SP | Υ | N | | Р | Υ | 09/08/2020 | Υ | N | 10/20/2022 | N |
| Himelhoch | Seth | Co-Investigator | DP | Υ | N | MD<br>MPH | Р | Υ | 07/18/2022 | Υ | N | 02/08/2021 | N |
| Khanal | Rebika | Recruitment | SP | Υ | N | | Р | Υ | 02/04/2022 | Υ | N | 02/08/2021 | N |
| Rush | Craig | Co-Investigator | DP | Υ | N | PhD | Р | Υ | 10/29/2020 | Υ | N | 01/04/2021 | N |
| Thornton | Alice | Co-Investigator | SP | N | N | MD | Р | Υ | 04/06/2022 | Υ | N | 01/04/2021 | N |
| Wesley | Michael | Co-Investigator | SP | Υ | N | PhD | Р | Υ | 10/13/2020 | Υ | N | 02/05/2021 | N |
| Burris | Jessica | Recruitment | SP | Υ | N | | Р | Υ | 03/06/2020 | Υ | Υ | 04/25/2021 | N |
| Christian | Amy | Recruitment | SP | Υ | N | | Р | Υ | 07/22/2021 | Υ | Υ | 04/25/2021 | N |
| Jasinski | Lindsey | Co-Investigator | SP | Υ | N | PhD | Р | Υ | 08/05/2020 | Υ | Υ | 10/19/2022 | N |
| Kahl | Joan | Recruitment | SP | Υ | N | | Р | Υ | 11/02/2020 | Υ | Υ | 04/25/2021 | N |
| Sabitus | Kathryn | Consultant/Advisor | SP | Υ | N | | Р | Υ | 06/21/2022 | Υ | Υ | 10/20/2022 | N |
| Su | Amanda | Data Collection | SP | Υ | N | | Р | Υ | 06/02/2021 | | Υ | 10/20/2022 | N |

#### RESEARCH DESCRIPTION

0 unresolved comment(s)

You may attach a sponsor's protocol pages in the "Additional Information" section and refer to them where necessary in the Research Description. However, each prompt that applies to your study should contain at least a summary paragraph.

#### Pro Tips:

- Save your work often to avoid losing data.
- Use one of the attachment buttons in this section or under the Additional Information section to include supplemental
  information with your application. During the document upload process, you will be able to provide a brief description
  of the attachment.

#### **Background**

Include a brief review of existing literature in the area of your research. You should identify gaps in knowledge that should be addressed and explain how your research will address those gaps or contribute to existing knowledge in this area. For interventional research, search PubMed and ClinicalTrials.gov for duplicative ongoing and completed trials with same condition and intervention(s).

Importance of the Problem to Be Addressed. The proposed pilot study seeks to explore modulation of attentional bias and tobacco craving in PLWHA with one session of adequately dosed theta burst stimulation (TBS). Results of this trial will spur clinical research to further investigate the use of TBS as an adjunctive smoking cessation aid for PLWHA and could have broad implications for smoking cessation programs. Data obtained from this pilot study will also facilitate resubmission of a grant application examining adjunctive theta burst stimulation (TBS) combined with varenicline for smoking cessation in PLWHA. People living with HIV/AIDS (PLWHA) smoke at nearly three times the rate of the general population (1-7). These extraordinary smoking rates are associated with greater AIDS-related morbidity (8-10), non-AIDS related morbidity including non-AIDS-defining cancer, cardiovascular disease, pulmonary disease (11-18), and mortality (19-22). Smoking significantly impacts the progression and outcome of HIV disease and has been identified as the leading contributor to premature mortality in PLWHA (23). One study estimated PLWHA lose more years from smoking than from HIV infection (21). In our view, shared by others in the field, the single greatest health behavior change that could improve mortality is to assist smokers living with HIV/AIDS to quit smoking (23-30).

Pharmacotherapies for Smoking Cessation in PLWHA. Trials involving use of nicotine replacement therapy (NRT) have shown no effect on cessation rates when used alone (31, 32) and mild efficacy when used in combination with behavioral therapies in PLWHA (33-35). Adherence to NRT was also low (34). No controlled trials have compared NRT with other smoking cessation interventions in PLWHA (36). Although bupropion has been approved for smoking cessation in healthy adults, no randomized trials have explicitly examined the efficacy of bupropion for smoking cessation in PLWHA (36). There have also been concerns regarding interactions between bupropion and antiretroviral therapy (HAART)(37, 38). Varenicline is considered the most effective pharmacologic agent available for smoking cessation (39). There are no reported pharmacodynamic interactions between varenicline and HAART (37, 40). Varenicline was found to be safe and well tolerated for smoking cessation interventions among PLWHA (40-42). It showed higher continuous abstinence rates (OR=4.65, CI 1.71-12.67, p=0.003) compared to placebo during weeks 9-12 (43), when dosed for 12 weeks. In another trial combining varenicline and NRT resulted in significantly higher continuous abstinence at weeks 12 (OR=1.85, p=0.007) and 24 (OR=1.98, p=0.004) (44). Despite these results, suboptimal adherence to varenicline poses a significant barrier resulting in lower quit rates in community studies compared to clinical trials (45). The extant literature suggests the efficacy of pharmacotherapeutics prescribed as smoking cessations aids is suboptimal in smokers in general and PLWHA in particular (30, 36). These findings along with high smoking rates in PLWHA underscore the urgent need to identify novel adjuncts to augment the efficacy and sustainability of commonly prescribed pharmacotherapies for smoking cessation.

Transcranial magnetic stimulation (TMS). TMS is a form of noninvasive brain stimulation. TMS uses a magnetic field to generate tiny modulated doses of electric current at a focal brain site, leading to neural changes and consequently changes in behavior and illness symptoms (46). In psychiatric illnesses like major depressive disorder (MDD) and schizophrenia, TMS has been used to augment medication treatments or treat residual symptoms, which are addressed sub-optimally by pharmacotherapy (47, 48). TMS has revolutionized the treatment of major depressive disorder (MDD), leading to FDA approval in 2008 for 10 Hz protocol. Neuroimaging studies have shown neural effects from TMS to result from activity modulation at stimulation site and downstream effects at other brain regions (49). These downstream effects result from connectivity changes in networks involving proximal cortical stimulation target and distal network structures (49). TMS is safe and has been refined significantly over the last 20 years.

The neurobiology of nicotine addiction encompasses increased dopaminergic activity in the mesolimbic reward pathway (nucleus accumbens and ventral tegmental area), via removal of inhibitory GABAergic activity (50). TMS at the left dorsolateral prefrontal cortex (DLPFC) causes increased dopaminergic release at the site of application and downstream dopaminergic modulation in the reward pathway, consequently leading to reduced craving (51). A recent meta-analysis showed excitatory TMS to the left dorsolateral prefrontal cortex (DLPFC) showed a medium effect size for craving reduction for nicotine (Hedges' g 0.471, CI 0.820 to 0.122, p=0.008) (52). Importantly, across substances, including nicotine, number of stimulation pulses predicted the effect size for reductions in craving (52). TMS has been used for smoking cessation in a few clinical studies with otherwise healthy individuals (53). Ten previous studies have applied excitatory TMS (10-20 Hz), one study applied inhibitory TMS (1 Hz) and one previous study applied TBS to reduce craving for cigarettes in subjects with no comorbid psychiatric diagnoses (53). Number of sessions ranged from one to ten, with four being median (53). Eight studies targeted left or right DLPFC, one used an H coil targeting bilateral DLPFC and insula (54) and one study targeted the left superior frontal gyrus (55). Nine out of ten studies used craving measures as outcomes, all assessed abstinence from smoking cigarettes at various time points. All these have been pilot studies, with sample sizes ranging from 16 to 48.

Theta burst stimulation (TBS). A new TMS paradigm, theta burst stimulation (TBS), uses theta frequency stimulatid gamma frequency. TBS is different from other TMS frequencies in that it delivers significantly more dosing pulses over the same time period. TBS is safe and was approved for MDD by the FDA in 2019. To the best of our knowledge, there has been only a single clinical study that utilized theta burst stimulation for smoking cessation. Four sessions of intermittent TBS (iTBS) added to Cognitive Behavioral Therapy (CBT, twice weekly sessions for three weeks) (56) were delivered. Participants (N=74) received either iTBS (600 pulses) or sham TMS. The groups did not differ in number of cigarettes smoked or scores on Fagerstrom Test for Nicotine Dependence (FTND). At three months of follow-up, the iTBS group had 19 subjects reporting abstinence while 19 had relapsed. The sham TMS group had 10 subjects abstinent and 26 subjects who had relapsed. To the best of our knowledge, no studies used TBS or other rTMS for smoking cessation in PLWHA.

TMS for modulation of cognitive performance including attentional bias. TMS has also been used to modulate cognitive performance, to accelerate mechanisms of smoking cessation across various studies (57, 58). Previous TMS treatment studies for smoking cessation have included cognitive outcome measures including delayed discounting (59, 60) and cigarette cue induced craving assessed using an analogue scale (61). It is plausible modulation of these cognitive paradigms by TMS could contribute to craving reduction and behavioral changes in cigarette use. Multiple previous studies support the existence of an attentional bias towards smoking related cues compared to neutral cues in tobacco use disorder(62). Modulation of attentional bias has been attempted in MDD. To the best of our knowledge, no study has used TMS to modulate attentional bias in subjects with smoking behavior.

Stress induced craving paradigm. The pathophysiology of nicotine dependence includes the interaction between stress, environment and body physiology, fuelling the illness(63). Multiple previous studies have modeled craving for nicotine in the presence of stress, to approximate real world scenarios(64-66). Before we test TBS as a clinical intervention, we will explore whether one session of TBS can modulate craving in the context of induced stress. Two promising paradigms for stress induction are the cold pressor test (CPT) wherein participants immerse their feet in ice cold water (2-4 degree Celsius) for three minutes and the paced serial addition task (PASAT)(67). The cold pressor test invokes an immediate cardiovascular stress response, initiated by the sympathetic nervous system, followed by a neuroendocrine response controlled by the hypothalamus-pituitary-adrenal (HPA) axis(67). The PASAT is a cognitively challenging task and will be performed in parallel with the CPT as an additional means for stress induction. The task requires participants to listen to a standardized audio-recording of a series of single-digit numbers and to say aloud the sum of the last two numbers presented (within each inter-trial interval). The PASAT will also last less than three minutes. Peak stress response occurred 20 minutes after these paradigms were performed(67). In our pilot study, these paradigms will be performed simultaneously, and followed by the tobacco craving questionnaire (TCQ).

Brain network connectivity to complement attentional bias modulation. Neuroimaging has shown resting state functional connectivity (rsFC) changes in patients who smoke(68). This encompasses connectivity changes in default mode network, executive control network and salience network. Previous studies have shown a negative correlation between smoking behavior severity and connectivity in the dorsal anterior cingulate (dACC)- ventral striatum (VS) circuit(68). Previous studies have also shown the salience network to be deeply involved in the regulation of attention to smoking cues versus neutral cues(68). Given that neuroimaging could potentially corroborate attentional bias modulation with TBS, we will attempt to explore correlations between changes in attentional bias and salience network as well as between changes in stress induced craving and connectivity in the dACC-VS circuit.

#### References

- 1. Kwong J, Bouchard-Miller K, Smoking cessation for persons living with HIV: a review of currently available interventions. J Assoc Nurses AIDS Care, 2010;21(1):3-10.
- 2. Niaura R, Shadel WG, Morrow K, Tashima K, Flanigan T, Abrams DB. Human immunodeficiency virus infection, AIDS, and smoking cessation: the time is now. Clin Infect Dis. 2000;31(3):808-12.
- 3. Tesoriero JM, Gieryic SM, Carrascal A, Lavigne HE. Smoking among HIV positive New Yorkers: prevalence, frequency, and opportunities for cessation. AIDS Behav. 2010;14(4):824-35.
- 4. Burkhalter JE, Springer CM, Chhabra R, Ostroff JS, Rapkin BD. Tobacco use and readiness to quit smoking in low-income HIV-infected persons. Nicotine Tob Res. 2005;7(4):511-22.
- 5. Moscou-Jackson G, Commodore-Mensah Y, Farley J, Digiacomo M. Smoking-Cessation Interventions in People Living With HIV Infection: A Systematic Review. J Assoc Nurses AIDS Care. 2013.
- 6. Lifson AR, Lando HA. Smoking and HIV: prevalence, health risks, and cessation strategies. Curr HIV/AIDS Rep. 2012;9(3):223-30.
- 7. Mamary EM, Bahrs D, Martinez S. Cigarette smoking and the desire to quit among individuals living with HIV. AIDS Patient Care STDS. 2002;16(1):39-42.
- 8. Feldman JG, Minkoff H, Schneider MF, Gange SJ, Cohen M, Watts DH, et al. Association of cigarette smoking with HIV prognosis among women in the HAART era: a report from the women's interagency HIV study. Am J Public Health. 2006;96(6):1060-5.
- 9. Cropsey KL, Willig JH, Mugavero MJ, Crane HM, McCullumsmith C, Lawrence S, et al. Cigarette Smokers are Less Likely to Have Undetectable Viral Loads: Results From Four HIV Clinics. J Addict Med. 2016;10(1):13-9.
- 10. Nieman RB, Fleming J, Coker RJ, Harris JR, Mitchell DM. The effect of cigarette smoking on the development of AIDS in HIV-1-seropositive individuals. AIDS. 1993;7(5):705-10.
- 11. Metersky ML, Colt HG, Olson LK, Shanks TG. AIDS-related spontaneous pneumothorax. Risk factors and treatment. Chest. 1995;108(4):946-51.
- 12. Saves M, Chene G, Ducimetiere P, Leport C, Le MG, Amouyel P, et al. Risk factors for coronary heart disease in patients treated for human immunodeficiency virus infection compared with the general population. Clin Infect Dis. 2003;37(2):292-8.
- 13. Palella FJ, Jr., Phair JP. Cardiovascular disease in HIV infection. Curr Opin HIV AIDS. 2011;6(4):266-71.
- 14. Winstone TA, Man SF, Hull M, Montaner JS, Sin DD. Epidemic of lung cancer in patients with HIV infection. Chest. 2013;143(2):305-14.
- 15. De P, Farley A, Lindson N, Aveyard P. Systematic review and meta-analysis: influence of smoking cessation on incidence of pneumonia in HIV. BMC Med. 2013;11:15.
- 16. Akgun KM, Gordon K, Pisani M, Fried T, McGinnis KA, Tate JP, et al. Risk factors for hospitalization and medical intensive care unit

- (MICU) admission among HIV-infected Veterans, J Acquir Immune Defic Syndr, 2013;62(1):52-9,
- 17. Calvo-Sanchez M, Perello R, Perez I, Mateo MG, Junyent M, Laguno M, et al. Differences between HIV-infected and unintected adults in the contributions of smoking, diabetes and hypertension to acute coronary syndrome: two parallel case-control studies. HIV Med. 2013;14(1):40-8.
- 18. Kingsley LA, Deal J, Jacobson L, Budoff M, Witt M, Palella F, et al. Incidence and progression of coronary artery calcium in HIV-infected and HIV-uninfected men. AIDS. 2015;29(18):2427-34.
- 19. Crothers K, Goulet JL, Rodriguez-Barradas MC, Gibert CL, Oursler KA, Goetz MB, et al. Impact of cigarette smoking on mortality in HIV-positive and HIV-negative veterans. AIDS Educ Prev. 2009;21(3 Suppl):40-53.
- 20. Lifson AR, Neuhaus J, Arribas JR, Berg-Wolf M, Labriola AM, Read TR. Smoking-related health risks among persons with HIV in the Strategies for Management of Antiretroviral Therapy clinical trial. Am J Public Health. 2010;100(10):1896-903.
- 21. Helleberg M, May MT, Ingle SM, Dabis F, Reiss P, Fatkenheuer G, et al. Smoking and life expectancy among HIV-infected individuals on antiretroviral therapy in Europe and North America: The ART Cohort Collaboration. AIDS. 2014.
- 22. Morlat P, Roussillon C, Henard S, Salmon D, Bonnet F, Cacoub P, et al. Causes of death among HIV-infected patients in France in 2010 (national survey): trends since 2000. AIDS. 2014;28(8):1181-91.
- 23. Davies TL, Gompels M, Johnston S, Bovill B, May MT. Mind the gap: difference between Framingham heart age and real age increases with age in HIV-positive individuals-a clinical cohort study. BMJ Open. 2013;3(10):e003245.
- 24. Lundgren JD, Battegay M, Behrens G, de WS, Guaraldi G, Katlama C, et al. European AIDS Clinical Society (EACS) guidelines on the prevention and management of metabolic diseases in HIV. HIV Med. 2008;9(2):72-81.
- 25. Treating tobacco use and dependence: 2008 update U.S. Public Health Service Clinical Practice Guideline executive summary. Respir Care. 2008;53(9):1217-22.
- 26. Grinspoon SK, Grunfeld C, Kotler DP, Currier JS, Lundgren JD, Dube MP, et al. State of the science conference: Initiative to decrease cardiovascular risk and increase quality of care for patients living with HIV/AIDS: executive summary. Circulation. 2008;118(2):198-210.
- 27. Hoffman AC, Starks VL, Gritz ER. The impact of cigarette smoking on HIV/AIDS: urgent need for research and cessation treatment. AIDS Educ Prev. 2009;21(3 Suppl):1-2.
- 28. Nahvi S, Cooperman NA. Review: the need for smoking cessation among HIV-positive smokers. AIDS Educ Prev. 2009;21(3 Suppl):14-27.
- 29. Niaura R, Chander G, Hutton H, Stanton C. Interventions to address chronic disease and HIV: strategies to promote smoking cessation among HIV-infected individuals. Curr HIV/AIDS Rep. 2012;9(4):375-84.
- 30. Pacek LR, Cioe PA. Tobacco Use, Use Disorders, and Smoking Cessation Interventions in Persons Living With HIV. Curr HIV/AIDS Rep. 2015;12(4):413-20.
- 31. Moadel AB, Bernstein SL, Mermelstein RJ, Arnsten JH, Dolce EH, Shuter J. A randomized controlled trial of a tailored group smoking cessation intervention for HIV-infected smokers. J Acquir Immune Defic Syndr. 2012;61(2):208-15.
- 32. Shuter J, Morales DA, Considine-Dunn SE, An LC, Stanton CA. Feasibility and preliminary efficacy of a web-based smoking cessation intervention for HIV-infected smokers: a randomized controlled trial. J Acquir Immune Defic Syndr. 2014;67(1):59-66.
- 33. Stanton CA, Papandonatos GD, Shuter J, Bicki A, Lloyd-Richardson EE, de Dios MA, et al. Outcomes of a Tailored Intervention for Cigarette Smoking Cessation Among Latinos Living With HIV/AIDS. Nicotine Tob Res. 2015;17(8):975-82.
- 34. Ingersoll KS, Cropsey KL, Heckman CJ. A test of motivational plus nicotine replacement interventions for HIV positive smokers. AIDS Behav. 2009;13(3):545-54.
- 35. Lloyd-Richardson EE, Stanton CA, Papandonatos GD, Shadel WG, Stein M, Tashima K, et al. Motivation and patch treatment for HIV+ smokers: a randomized controlled trial. Addiction. 2009;104(11):1891-900.
- 36. Ledgerwood DM, Yskes R. Smoking Cessation for People Living With HIV/AIDS: A Literature Review and Synthesis. Nicotine Tob Res. 2016;18(12):2177-84.
- 37. Park-Wyllie LY, Antoniou T. Concurrent use of bupropion with CYP2B6 inhibitors, nelfinavir, ritonavir and efavirenz: a case series. AIDS. 2003;17(4):638-40.
- 38. Hesse LM, Greenblatt DJ, von Moltke LL, Court MH. Ritonavir has minimal impact on the pharmacokinetic disposition of a single dose of bupropion administered to human volunteers. J Clin Pharmacol. 2006;46(5):567-76.
- 39. Gibbons RD, Mann JJ. Varenicline, smoking cessation, and neuropsychiatric adverse events. Am J Psychiatry. 2013;170(12):1460-7.
- 40. Cui Q, Robinson L, Elston D, Smaill F, Cohen J, Quan C, et al. Safety and tolerability of varenicline tartrate (Champix((R))/Chantix((R))) for smoking cessation in HIV-infected subjects: a pilot open-label study. AIDS Patient Care STDS. 2012;26(1):12-9.
- 41. Tornero C, Mafe C. Varenicline and antiretroviral therapy in patients with HIV. J Acquir Immune Defic Syndr. 2009;52(5):656.
- 42. Ferketich AK, Diaz P, Browning KK, Lu B, Koletar SL, Reynolds NR, et al. Safety of varenicline among smokers enrolled in the lung HIV study. Nicotine Tob Res. 2013;15(1):247-54.
- 43. Ashare RL, Thompson M, Serrano K, Leone F, Metzger D, Frank I, et al. Placebo-controlled randomized clinical trial testing the efficacy and safety of varenicline for smokers with HIV. Drug Alcohol Depend. 2019;200:26-33.
- 44. Pacek LR, McClernon FJ, Bosworth HB. Adherence to Pharmacological Smoking Cessation Interventions: A Literature Review and Synthesis of Correlates and Barriers. Nicotine Tob Res. 2018;20(10):1163-72.
- 45. Slotema CW, Blom JD, Hoek HW, Sommer IE. Should we expand the toolbox of psychiatric treatment methods to include Repetitive Transcranial Magnetic Stimulation (rTMS)? A meta-analysis of the efficacy of rTMS in psychiatric disorders. J Clin Psychiatry. 2010;71(7):873-84.
- 46. Petrides G, Malur C, Braga RJ, Bailine SH, Schooler NR, Malhotra AK, et al. Electroconvulsive therapy augmentation in clozapine-resistant schizophrenia: a prospective, randomized study. Am J Psychiatry. 2015;172(1):52-8.
- 47. Ward HB, Szabo ST, Rakesh G. Maintenance ECT in schizophrenia: A systematic review. Psychiatry Res. 2018;264:131-42.
- 48. Castrillon G, Sollmann N, Kurcyus K, Razi A, Krieg SM, Riedl V. The physiological effects of noninvasive brain stimulation fundamentally differ across the human cortex. Sci Adv. 2020;6(5):eaay2739.
- 49. Laviolette SR, van der Kooy D. The neurobiology of nicotine addiction: bridging the gap from molecules to behaviour. Nat Rev Neurosci. 2004;5(1):55-65.
- 50. Strafella AP, Paus T, Barrett J, Dagher A. Repetitive transcranial magnetic stimulation of the human prefrontal cortex induces

dopamine release in the caudate nucleus, J Neurosci, 2001;21(15):RC157,

- 51. Zhang JJQ, Fong KNK, Ouyang RG, Siu AMH, Kranz GS. Effects of repetitive transcranial magnetic stimulation (rTMS) on craving and substance consumption in patients with substance dependence: a systematic review and meta-analysis. Addiction. 2019.
- 52. Hauer L, Scarano Gl, Brigo F, Golaszewski S, Lochner P, Trinka E, et al. Effects of repetitive transcranial magnetic stimulation on nicotine consumption and craving: A systematic review. Psychiatry Res. 2019;281:112562.
- 53. Dinur-Klein L, Dannon P, Hadar A, Rosenberg O, Roth Y, Kotler M, et al. Smoking cessation induced by deep repetitive transcranial magnetic stimulation of the prefrontal and insular cortices: a prospective, randomized controlled trial. Biol Psychiatry. 2014;76(9):742-9.
- 54. Rose JE, McClernon FJ, Froeliger B, Behm FM, Preud'homme X, Krystal AD. Repetitive transcranial magnetic stimulation of the superior frontal gyrus modulates craving for cigarettes, Biol Psychiatry, 2011;70(8):794-9.
- 55. Dieler AC, Dresler T, Joachim K, Deckert J, Herrmann MJ, Fallgatter AJ. Can intermittent theta burst stimulation as add-on to psychotherapy improve nicotine abstinence? Results from a pilot study. Eur Addict Res. 2014;20(5):248-53.
- 56. Beynel L, Appelbaum LG, Luber B, Crowell CA, Hilbig SA, Lim W, et al. Effects of online repetitive transcranial magnetic stimulation (rTMS) on cognitive processing: A meta-analysis and recommendations for future studies. Neurosci Biobehav Rev. 2019;107:47-58.
- 57. Coles AS, Kozak K, George TP. A review of brain stimulation methods to treat substance use disorders. Am J Addict. 2018;27(2):71-91.
- 58. Sheffer CE, Bickel WK, Brandon TH, Franck CT, Deen D, Panissidi L, et al. Preventing relapse to smoking with transcranial magnetic stimulation: Feasibility and potential efficacy. Drug Alcohol Depend. 2018;182:8-18.
- 59. Sheffer CE, Mennemeier M, Landes RD, Bickel WK, Brackman S, Dornhoffer J, et al. Neuromodulation of delay discounting, the reflection effect, and cigarette consumption. J Subst Abuse Treat. 2013;45(2):206-14.
- 60. Pripfl J, Tomova L, Riecansky I, Lamm C. Transcranial magnetic stimulation of the left dorsolateral prefrontal cortex decreases cue-induced nicotine craving and EEG delta power. Brain Stimul. 2014;7(2):226-33.
- 61. Robinson JD, Versace F, Engelmann JM, Cui Y, Gilbert DG, Waters AJ, et al. Attentional bias to smoking and other motivationally relevant cues is affected by nicotine exposure and dose expectancy. J Psychopharmacol. 2016;30(7):627-40.
- 62. Field M, Cox WM. Attentional bias in addictive behaviors: a review of its development, causes, and consequences. Drug Alcohol Depend. 2008;97(1-2):1-20.
- 63. Coskunpinar A, Cyders MA. Impulsivity and substance-related attentional bias: a meta-analytic review. Drug Alcohol Depend. 2013;133(1):1-14.
- 64. Sinha R. Modeling stress and drug craving in the laboratory: implications for addiction treatment development. Addict Biol. 2009;14(1):84-98.
- 65. McKee SA, Sinha R, Weinberger AH, Sofuoglu M, Harrison EL, Lavery M, et al. Stress decreases the ability to resist smoking and potentiates smoking intensity and reward. J Psychopharmacol. 2011;25(4):490-502.
- 66. Verplaetse TL, Weinberger AH, Oberleitner LM, Smith KM, Pittman BP, Shi JM, et al. Effect of doxazosin on stress reactivity and the ability to resist smoking. J Psychopharmacol. 2017;31(7):830-40.
- 67. Kotlyar M, Drone D, Thuras P, Hatsukami DK, Brauer L, Adson DE, et al. Effect of stress and bupropion on craving, withdrawal symptoms, and mood in smokers. Nicotine Tob Res. 2011;13(6):492-7.
- 68. Bachmann P, Finke JB, Rebeck D, Zhang X, Larra MF, Koch KP, et al. Test-retest reproducibility of a combined physical and cognitive stressor. Biol Psychol. 2019;148:107729.
- 69. Fedota JR, Stein EA. Resting-state functional connectivity and nicotine addiction: prospects for biomarker development. Ann N Y Acad Sci. 2015;1349:64-82.
- 70. Suppa A, Huang YZ, Funke K, Ridding MC, Cheeran B, Di Lazzaro V, et al. Ten Years of Theta Burst Stimulation in Humans: Established Knowledge, Unknowns and Prospects. Brain Stimul. 2016;9(3):323-35.
- 71. Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, et al. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020;177(8):716-26.
- 72. Heishman SJ, Singleton EG, Pickworth WB. Reliability and validity of a Short Form of the Tobacco Craving Questionnaire. Nicotine Tob Res. 2008;10(4):643-51.
- 73. Ekhtiari H, Kuplicki R, Pruthi A, Paulus M. Methamphetamine and Opioid Cue Database (MOCD): Development and Validation. Drug Alcohol Depend. 2020;209:107941.
- 74. Alcorn JL, 3rd, Strickland JC, Lile JA, Stoops WW, Rush CR. Acute methylphenidate administration reduces cocaine-cue attentional bias. Prog Neuropsychopharmacol Biol Psychiatry. 2020;103:109974.

### **Objectives**

List your research objectives. Please include a summary of intended research objectives in the box below.

Before the study proper, we will conduct a pilot study to validate our attentional bias task in healthy controls who may or may not have a history of current or active smoking. The specific aim of this pilot would be to show differences in attentional bias between smokers and non smokers.

Study proper. Specific Aim 1 will demonstrate whether one session of MRI targeted TBS to left dorsolateral prefrontal cortex (DLPFC) will decrease attentional bias to smoking cues, compared to sham TMS. Subjects will receive both one TBS session (1800 pulses) and one session of sham TMS, lasting 10 minutes on separate days. They will perform an attentional bias task before and after TBS. We hypothesize that TBS will significantly decrease post session attentional bias to smoking cues compared to sham TMS. Specific Aim 2 will demonstrate whether one session of TBS versus sham TMS, to left DLPFC can modulate stress induced craving for smoking. Subjects will perform the short form of tobacco craving questionnaire (TCQ-SF) before and after TBS. We hypothesize TBS will significantly decrease craving in smoking patients compared to sham TMS.

Specific Aim 3 will demonstrate whether one session of TBS versus sham TMS, to left DLPFC can increase seed based functional connectivity (fc) in the ventral striatum. We will acquire resting state functional MRI (fMRI) scans before and after TBS in all subjects. We hypothesize increase in fc in the dorsal anterior cinqulate – ventral striatum circuit after TBS.

### Study Design

Describe and explain the study design (e.g., observational, secondary analysis, single/double blind, parallel, crossover, deception, etc.).

- Clinical Research: Indicate whether subjects will be randomized and whether subjects will receive any placebo.
- Community-Based Participatory Research: If you are conducting <u>community-based participatory research (CBPR)</u>, describe strategies for involvement of community members in the design and implementation of the study, and dissemination of results from the study.
- Qualitative research: Indicate ranges where flexibility is needed, if a fixed interview transcript is not available, describe interview
  topics including the most sensitive potential questions.
- Research Repositories: If the purpose of this submission is to establish a Research Repository (bank, registry) and the material
  you plan to collect is already available from a commercial supplier, clinical lab, or established IRB approved research repository,
  provide scientific justification for establishing an additional repository collecting duplicate material. Describe the repository design
  and operating procedures. For relevant information to include, see the <u>UK Research Biospecimen Bank Guidance</u> or the <u>UK
  Research Registry Guidance</u>.

Before the actual study, we will conduct a pilot study involving 30 healthy controls who may or may not have a history of current or active smoking. They will perform the attentional bias task that we plan to use in the study proper. This would be an open label study, each subject would perform two versions of the attentional bias task lasting close to a total of 30 minutes.

Study Proper. This will be a double blind randomized controlled trial. All subjects will receive both TBS and sham TMS in a randomized manner with counter balancing. The TBS session and sham TMS will be done on separate days. Subjects will be randomized to receive either TBS first and sham TMS second, or sham TMS first and TBS second. The PI (Dr Rakesh) will be blind to the randomization status and will supervise the TMS session. Subjects will also remain blind to the randomization status. This will be facilitated by the Magventure Active/sham TMS coil which has been shown to maintain integrity of blinding in subjects regarding group assignment. We will recruit 30 patients from one of these clinics - the Bluegrass Clinic, SMART clinic in psychiatry and Beyond Birth Clinic in Psychiatry. All of them would receive TBS and sham TMS on separate days. The Bluegrass HIV clinic has a closely monitored population of PLWHA patients. The PI (Rakesh) and a research assistant would interface with Dr Alice Thornton at the Bluegrass HIV Clinic on a weekly basis and with Katie Sabitus on a daily basis to recruit patients for this study. The PI (Rakesh) and the research assistant will also interface with Dr Lindsey Jasinski (who heads the SMART clinic and Beyond Birth Clinic) on a weekly basis. If interested in participating, we will provide subjects with information and seek informed consent before proceeding with the study.

A sequential timeline of assessments and interventions are shown in table one. After informed consent, subjects will get an MRI brain scan at the Magnetic Resonance Imaging and Spectroscopy Center (MRISC) affiliated with University of Kentucky. Subjects will also be escorted to the MRISC at the UK Medical Center by the PI (Rakesh) and a research assistant. Subsequently, neuroimaging data (MRI brain) will be acquired using a Siemens 3-Tesla (3T) PRISMA MRI scanner as described under Data Collection below. This will happen on day 1. Then, on days 2 and 3, subjects will be scheduled for three hour experimental sessions at the TMS Suite at 245 Fountain Court, Lexington 40509. During these three hour sessions, subjects will perform the tobacco craving questionnaire (TCQ) while performing stress induced craving paradigm, attentional bias task and delayed discounting task. These activities will last an hour. Then we will obtain active motor threshold (AMT) from the first dorsal interosseous (FDI) muscle and left motor cortex, following which we will administer either a session of theta burst stimulation (TBS) for 9 minutes at 80% active motor threshold (AMT) or sham TMS to the left dorsolateral prefrontal cortex using a figure 8 coil and MagVenture MagPro x100 device (MagVenture A/S, Denmark), with TMS coil position stabilized using BrainSight (Rogue Solutions, Montreal, Canada). We will record motor evoked potential before and after the TBS session to assess response (10% increase in MEP to be a cutoff parameter). These activities will last another hour. After the TBS/sham TMS session, subjects will perform TCQ concomitant with the stress induced craving paradigm, attentional bias and delayed discounting tasks. These will last an hour. Then subjects will be transported to MRISC for their post TBS session MRI brain scan in the 3-Tesla (3T) PRISMA scanner.

Table 1
Study Task Study Day Pre- TBS Post-TBS
Urine Pregnancy Test 1
MRI brain at MRISC (Pre-TBS) 1
Exhaled CO 2 and 3 X
Motor Threshold 2 and 3 X
Eye tracking to measure AB 2 and 3 X X
Delayed Discounting Task 2 and 3 X X
Tobacco Craving Questionnaire 2 and 3 X X
TMS Side Effects Questionnaire 2 and 3 X
Treatment Acceptability Questionnaire 2 and 3 X
MRI brain at MRISC (Post-TBS) 2 and 3 X

#### Attachments

#### **Subject Recruitment Methods & Advertising**

Describe how the study team will identify and recruit subjects. Please consider the following items and provide additional information as needed so that the IRB can follow each step of the recruitment process.

- How will the study team identify potential participants?
- Who will first contact the potential subjects, and how?
- Will you use advertisements? If so, how will you distribute those?

- How and where will the research team meet with potential participants?
- If applicable, describe proposed outreach programs for recruiting women, minorities, or disparate populations.
- How you will minimize undue influence in recruitment?
- Attach copies of all recruiting and advertising materials (emails, verbal scripts, flyers, posts, messages, etc.).

For additional information on recruiting and advertising:

- IRB Application Instructions Advertisements
- PI Guide to Identification and Recruitment of Human Subjects for Research

For the pilot study, we will recruit 30 healthy volunteer subjects from in and around 245 Fountain Court to perform the computer based attentional bias task. This would essentially comprise office staff and other employees in 245 Fountain Court. There will be no coercion and subjects can individually choose if they would like to participate in this pilot study. Each subject would be administered two versions of the task for a total of approximately 30 minutes.

For the study proper, we will recruit 30 subjects from the Bluegrass HIV Clinic, SMART clinic and Beyond Birth Clinic. Study members will interface with all providers in these clinics on a daily basis. All providers in these clinics will be provided multiple copies of the study flyer. All providers in these clinics will also be informed about inclusion and exclusion criteria for the study, based on which all patients will be screened by them. The PI (Dr Rakesh) and a research assistant will interface with a contact in each of these clinics on a daily basis. Business cards (that list a few study details and a call back number if subjects are interested in the study) will be provided to subjects at each of these clinics by clinic providers. The case manager for this clinic Robert Bell will send an email to all patients from the clinic, with the study flyer attached and informing them about the study. Subjects interested in the study can call the number provided on the business card to express interest in the study. This number belongs to the PI (Dr Rakesh). He or the research assistant will administer a phone script to subjects who call back to assess subjects' suitability for the study. Once a subject is identified as suitable for the study, they will be asked to meet Dr Rakesh/research assistant at 245 Fountain Court to get informed consent if they are interested in study participation and fulfill other eligibility criteria for the study. This process will also encompass MRI screening, examining urine drug screen and breathalyzer results. Following this step, patients will be randomized to either the treatment arm or sham arm by study co-investigator Craig Rush. Half of compensation for study participation would be provided prior to starting the study and rest of it at study completion. All data collected from phone screening would be entered into RedCap, regardless of whether subjects do or don't fulfill inclusion and exclusion criteria.

Pertaining to the modification of study design - For subjects who have already participated in our trial and received one TMS session, we will inform them about this modification and ask them if they would be interested in coming back to receive another session of TMS (which may be active or sham, they will receive the opposite of what they got initially). The randomization procedure will be supervised by Dr Craig Rush this will be factored into the randomization counterbalancing procedure. We will educate participants who have completed the study previously on the modification of study design and offer them the modified consent form to read and sign if they are interested in participating in the third day of the study.

No flyers will be created for the pilot study. For the main study, we will create study flyers for providers at three clinics. These will list inclusion and exclusion criteria for the study as well as contact numbers for the PI (Gopalkumar Rakesh) and research assistant involved in the study.

#### Attachments

| Attach Type | ile Name |
|-------------|-----------------------------------------|
| Advertising | 64473_business_card PR edit STAMPED.pdf |
| Advertising | Bell_email.docx |
| Advertising | Rakesh_Flyer PR STAMPED.pdf |

#### **Research Procedures**

Describe how the research will be conducted.

- What experience will study participants have?
- What will study participants be expected to do?
- · How long will the study last?
- Outline the schedule and timing of study procedures.
- Provide visit-by-visit listing of all procedures that will take place.
- Identify all procedures that will be carried out with each group of participants.
- Describe deception and debrief procedures if deception is involved.

Differentiate between procedures that involve standard/routine clinical care and those that will be performed specifically for this research project. List medications that are explicitly forbidden or permitted during study participation.

Before the study proper, we will run a pilot to validate the attentional bias task. In this pilot, 20 subjects with current or previous history of smoking as well as 20 subjects with no history of current or previous smoking will perform a computerized behavioral task that examines attentional bias to smoking cues versus neutral cues. Subjects will perform the attentional bias task following informed consent. Following informed consent, they will undergo breathalyzer and CO estimation prior to the study session.

#### Study Proper

Following informed consent, the subject will be asked to come to MRISC for a MRI brain scan contingent on the investigative team obtaining a slot for this. The PI will coordinate with staff at MRISC to obtain a MRI slot. Subjects will also be escorted to the MRISC at the UK Medical Center by the PI (Rakesh) and a research assistant. Neuroimaging data (MRI brain) will be acquired using a Siemens 3-Tesla (3T) PRISMA scanner as described under Data Collection below. This will happen on day 1 and will last an hour. Then, on days 2 and 3, subjects will be scheduled for three hour experimental sessions at the TMS Suite at 245 Fountain Court, Lexington 40509. During these three hour sessions, subjects will perform the tobacco craving questionnaire (TCQ) while performing stress induced craving paradigm, attentional bias task and delayed discounting task. These activities will last an hour. Then we will obtain active motor threshold (AMT) from the first dorsal interosseous (FDI) muscle and left motor cortex, following which we will administer either a session of theta burst stimulation (TBS) for 9 minutes at 80% active motor threshold (AMT) or sham TMS to the left dorsolateral prefrontal cortex using a figure 8 coil and MagVenture MagPro x100 device (MagVenture A/S, Denmark), with TMS coil position stabilized using BrainSight (Rogue Solutions, Montreal, Canada). We will record motor evoked potential before and after the TBS session to assess response (10% increase in MEP to be a cutoff parameter). These activities will last another hour. After the TBS/sham TMS session, subjects will perform TCQ concomitant with the stress induced craving paradigm, attentional bias and delayed discounting tasks. These will last an hour. Then subjects will be transported to MRISC for their post TBS session MRI brain scan in the 3-Tesla (3T) PRISMA scanner.

#### Motor Threshold

Motor threshold (MT) is defined as the TMS pulse amplitude needed to elicit an EMG response of 50 µV peak-to-peak average amplitude in a target muscle. MT is the standard in the field for determining the intensity of TMS for everyone to reduce seizure risk. The MEP for the right first dorsal interosseus (FDI) will be measured with EMG. The scalp region producing the largest amplitude MEP will be identified. At that scalp location, we will determine the TMS intensity eliciting average MEP amplitude of 50 µV peak-to-peak in the first DI muscle using an amplitude titration procedure (at least 5/10 trials). Individual MT will be used to determine the intensity of theta burst stimulation for everyone, as recommended by safety guidelines.

### TBS application

A magnetic coil will be placed on the scalp and held in place with frameless stereotaxic equipment, using a sophisticated method of coil placement that will coregister scalp positions directly onto an average brain template. This Frameless Stereotaxic System Brainsight offers real-time three-dimensional display of cortical localization as the TMS coil is moved across the scalp. This will be used for coil positioning. This system uses a programmed robot arm to precisely position the TMS coil, and maintain its position, within 1 mm of the brain target chosen. Earplugs will be worn to protect hearing and low-volume white noise will be played through TMS-compatible headphones to mask the sound of the coil clicks. The intensity of the stimulation will be 120% of resting motor threshold as reported in a previous studies. The participant will be seated comfortably with headphones and earplugs to protect the subject's hearing. Before applying TBS or sham TMS, we provide subjects without scalp hair the option to apply 5% lidocaine spray (aspercreme) that is available over the counter to the left frontal quadrant of their scalp. This would minimize discomfort if any they feel during the stimulation. They would have the option to refuse as well.

### Stress induced craving paradigm

The pathophysiology of nicotine dependence includes the interaction between stress, environment and body physiology. Multiple previous studies have modeled craving for nicotine in the presence of stress, to approximate real world scenarios. Before we test TBS as a clinical intervention, we will explore whether one session of TBS can modulate craving in the context of induced stress. Two promising paradigms for stress induction are the cold pressor test (CPT) wherein participants immerse their feet in ice cold water (2-4 degree Celsius) for three minutes and the paced serial addition task (PASAT). The cold pressor test invokes an immediate cardiovascular stress response, initiated by the sympathetic nervous system, followed by a neuroendocrine response controlled by the hypothalamus-pituitary-adrenal (HPA) axis. The PASAT is a cognitively challenging task and will be performed in parallel with the CPT as an additional means for stress induction. The task requires participants to listen to a standardized audio-recording of a series of single-digit numbers and to say aloud the sum of the last two numbers presented (within each inter-trial interval). The PASAT will also last about three minutes. Peak stress response occurred 20 minutes after these paradigms were performed. In our pilot study, these paradigms will be performed simultaneously, and followed by the tobacco craving questionnaire (TCQ).

The Tobacco Craving Questionnaire-short form (TCQ-SF)

It consists of 12 items rated on a visual analogue scale. The original Tobacco Craving Questionnaire (TCQ) is a valid and reliable 47item self-report instrument that assesses tobacco craving in four dimensions: emotionality, expectancy, compulsivity, and purposefulness. The short form has been found to be as valid and reliable as the original version.

#### Attentional Bias task

We will measure attentional bias using a validated database of smoking and neutral cues and Tobii Pro Fusion 120 Hz eye tracker (Tobii Technology, Sweden). Smoking and neutral cues will be presented side-by-side on the screen for 1000?milliseconds. Eye tracking will record eye movements and fixation times for both cue types. Upon offset of the cues, a visual probe ('X') will appear on either the left or right side of the computer screen. Participants will be instructed to respond as quickly as possible to the probe. The primary dependent variable will be mean fixation time (milliseconds) calculated by summing the total fixation time for each cue type and then dividing by the total number of critical trials (i.e., 40). Reaction times to the visual probe will also be collected.

#### Attention bias behavioral activation (ABBA) task using go/no go

A modified cued go/no-go task is used as a measure of inhibitory control. The procedures and parameters for the attentional bias-behavioral activation (ABBA) task are identical to the traditional cued go/no-go task except that opiate-related images serve as go cues and neutral images serve as no-go cues. Opiate related images and neutral images that will be used for this task are attached below.

#### Delayed discounting task

Participants are presented a fixed set of 27 choices between smaller, immediate rewards (SIRs) and larger, delayed rewards (LDRs). Three trials of the task are presented, money versus money, money versus opiate reward, and opiate versus opiate reward in varying amounts and with varying time periods. The 27 choices in each of these trial types define ten ranges of discount rates, eight of which are bounded above and below and two of which represent the endpoints (choices of all 27 immediate rewards or all 27 delayed rewards). Based on participants' choices of the immediate reward across trials, each participant is assigned a k value corresponding to the geometric midpoint of one of the eight ranges or one of the two endpoint values. Each participant is assigned a k value that yields the highest proportion of choices consistent with that assignment. That is, for each participant we compute the proportion of that person's choices that were consistent with assignment to each of the 10 values of k defined by the questionnaire (bounded or unbounded), and the participant is assigned to the value that yields the highest consistency among his or her choices. The discount rate that yields the highest relative consistency across trials provides the best estimate of the participant's k value. When two or more values yielded equal consistency, the participant is assigned a value corresponding to the geometric mean of those values. The discounting rate (k) is estimated with nonlinear regression using Mazur's (1987) hyperbolic-decay model, vd = V/ (1+kd), where V is the value of a an outcome delayed by d days and vd is the value of the immediate outcome – a proportion of V subjectively discounted at "rate" k. Distributions of k-values transformed with the natural logarithm (In) tend to be approximately normal.

Barratt impulsiveness scale (BIS-11) - The BIS-11 is a 30-item self-report questionnaire to assess impulsivity that has been validated in multiple studies and other languages.

| Attack | ments |
|--------|-----------|
| Allaci | IIIIeiits |

| Attach Type | File Name |
|--------------------|-----------|
| ResearchProcedures | COC.pdf |

#### **Data Collection & Research Materials**

In this section, please provide the following:

- Describe all sources or methods for obtaining research materials about or from living individuals (such as specimens, records, surveys, interviews, participant observation, etc.), and explain why this information is needed to conduct the study.
- For each source or method described, please list or attach all data to be collected (such as genetic information, interview scripts, survey tools, data collection forms for existing data, etc.).
- If you will conduct a record or chart review, list the beginning and end dates of the records you will view.

Motor Threshold

Eve tracking

Delay discounting task

Attention bias behavioral activation (ABBA) task using go/no go

Barratt impulsiveness scale (BIS-11)

Tobacco Craving questionnaire (TCQ)

TMS Side effects scale

Treatment acceptability questionnaire (TAQ)

Resting state functional magnetic resonance imaging (fMRI)

Neuroimaging data will be acquired on a Siemens 3-Tesla (3T) PRISMA scanner. A high-resolution (1 cubic millimeter voxels) T1-weighted MP-RAGE structural image will be acquired for each subject. Functional images will be acquired using echo-planar imaging. Hyper-angulated volumes will be acquired with 37 ascending and interleaved slices at an angle 30-degrees to the anterior-posterior commissure to prevent OFC washout. Additional parameters will be similar to those used in other approved neuroimaging protocols in our lab (e.g., a repetition time (TR) of 2 seconds, echo time (TE) of 25 ms, a flip angle of 90 degrees, and functional voxels of size 3.4mm x 4.0mm). Image preprocessing will be performed in statistical parametric mapping (SPM) 12 software using standard procedures (see Wesley et al., 2014). Data from functional scans will be treated similarly to fMRI data in previous studies

(e.g., slice-timing corrected, head-motion corrected, warped into MNI standard space, re-sliced to 4 cubic millimet smoothed with an 8mm full-width, half-maximum (FWHM) Gaussian kernel).

### Attachments

| Attach Type | File Name |
|----------------|-----------------------------------------|
| DataCollection | PreScrnF.pdf |
| DataCollection | entional_Bias_Behavioral_Activation.pdf |
| DataCollection | BIS.pdf |
| DataCollection | Stress paradigms.pdf |
| DataCollection | TCQ-SF.png |
| DataCollection | TMS_Side effects.doc |
| DataCollection | TAQ.PNG |
| DataCollection | Delayed_discounting choices.docx |

#### Resources

Describe the availability of the resources and adequacy of the facilities that you will use to perform the research. Such resources may include:

- Staffing and personnel, in terms of availability, number, expertise, and experience;
- Computer or other technological resources, mobile or otherwise, required or created during the conduct of the research;
- Psychological, social, or medical services, including equipment needed to protect subjects, medical monitoring, ancillary care, or counseling or social support services that may be required because of research participation;
- Resources for communication with subjects, such as language translation/interpretation services.

Personnel: PI (Gopalkumar Rakesh), Co-Investigators (Seth Himelhoch, Craig Rush, Michael Wesley, Lindsey Jasinski), research Assistant,

The TMS Suite is housed within the department of psychiatry (245 Fountain Court, Lexington, Kentucky 40509) at the University of Kentucky, Lexington. Currently it encompasses one experimental room covering about 600 sq feet on the second floor. We are in the process of purchasing a a MagPro X100 stimulator (MagVenture Inc, Atlanta,GA) with booster option and active cooling. The room will also also equipped with a laptop and a chair to provide TMS. The device is capable of producing rTMS over a wide range of parameters such as paired-pulse, theta burst stimulation, and both monophasic and biphasic waveforms. The machine weighs 35 kg and the cart encompassing the machine weighs 16 kg. Dimensions of the machine are 210 x 530 x 400 mm. We are also in the process of purchasing a frameless stereotaxic system (Brainsight Frameless, Rogue Research, Montreal, QC, Canada) for coregistration of TMS coil position on the scalp with underlying cortical anatomy on the individual subject's three-dimensionally rendered MRI scan. This permits navigation of the TMS coil to target cortical structures. Participants are administered TMS in a customized chair for stabilization of head and coil position. A coil holder especially designed for TMS ensures stable coil positioning. The Brainsight Neuronavigation system has three main components: (1) NDI Spectra infrared camera system, (2) stimulator, (3) chair with neck rest. The TMS coil is targeted to a user defined location selected on the individual 3-D Anatomical MRI with fMRI or PET data overlay with less than one millimeter error. The TMS coil is attached to a stimulator unit, which administers the TMS pulses to modulate brain function in a spatially and temporally precise fashion. The subject reclines in the chair and wears a headband equipped with a subject position tracker. The ceiling mounted infrared stereo camera detects the 3-D position of the subject tracker and also the coil position tracker, and continuously feeds this information into the control center software.

Eye Tracker. The Tobii Pro Fusion housed at 245 Fountain Court is an exceptionally flexible remote eye tracking system offering supreme tracking performance in a wide array of human behavior research studies. This small eye tracking research system offers unprecedented portability and freedom of head movement in combination with unparalleled tracking accuracy and robust participant tracking capability. It allows for both screen and real-world test scenarios. For screen based research, it can be used with a laptop, an external monitor or an all-in-one PC. It can be mounted below most screens, With the eye tracker flush mounted on a screen, researchers can achieve highly accurate results for stimuli presentation on screens. Using a desk stand, one can track larger screens. This gives researchers the freedom to present stimuli on a screen that best meets the specific needs of the study at hand. The eye tracking system captures data up to speeds of 250 Hz (available 60, 120, 250 Hz modes). It delivers unparalleled data accuracy within the whole tracking box and very robust participant tracking capability. Robust eye tracking capability ensures very low data loss in real life conditions. The system with automatic selection of bright or dark pupil eye tracking accommodates for large variations in experimental conditions and demographic populations. The system also comes fitted with Tobii Pro Lab. This is a versatile biometric software platform designed for extensive research into human behavior using eye tracking analysis. It also has added ability to be combined with other physiological data streams. From in-store shopper research to psychology experiments, Pro Lab makes it easy for anyone to start using various biometric tools in their research in order to further expand the scope and richness of their insights. Pro Lab works well with both screen-based and wearable eye trackers.

Magnetic Resonance Imaging and Spectroscopy Center (MRISC). The Magnetic Resonance Imaging and Spectroscopy Center (MRISC) is a service and consultation center supporting basic and clinical research at the University of Kentucky. The Center includes an advanced 3T Siemens PRISMA scanner with high performance gradients, echo-planar whole body imaging and hydrogen spectroscopic capabilities for both human and animal studies. For dedicated animal studies, a modern Bruker/Siemens 7T MR scanner has recently been installed. Recently renovated facilities for animal handling, preparation and care are available immediately adjacent to the 7T imager. There are also computing facilities, electronic and fabrication shops, and a multi-user laboratory available to support magnetic resonance and spectroscopy studies. Scientific and technical personnel are available to help in developing MR

sequences and procedures as well as to help with image-processing analysis. The Center has multiple ongoing re https://www.research.uky.edu/magnetic-resonance-imaging-and-spectroscopy-center/human-research-projects.

In 2017 the MRISC was awarded an NIH grant to upgrade its human MRI scanner from a Siemens TIM TRIO 3T to a Siemens MAGNETOM Prisma 3T. The Prisma 3T offers maximum performance under prolonged high-strain conditions and delivers improved resolution over the previous system by coils with the highest gradient strength currently available on the market. Of note, data collected with the Prisma 3T scanner are to a higher-quality standard and are therefore more attractive for inclusion into NIH-supported neuroimaging repositories, such as the Neuroimaging Informatics Tools and Resources Clearinghouse (NITRC) and the Human Connectome Project (HCP). The Prisma 3T is equipped with a full complement of coils, updated image processing using Siemens Software 3D rendering, image fusion, perfusion, DTI fiber tracking, spectroscopy, volume rendering, shaded surface display, multiplanar reconstruction, and maximum intensity projection.

Ancillary Equipment in MRI Suite. 1) Applied Sciences Laboratories, Inc. Model 504LRO (long range optics) eye tracker complete with Real Eye software; 2) AVOTEC, Inc. Silent Vision SL-6011 LCD projection system used with Psychology Software Tools, Inc. visual presentation software, EPRIME; 3) MRA, Inc. 10 channel, fiber optic, patient response system with trigger interface and visual/auditory patient monitoring; 4) Current Designs, Inc. patient response fORP Interface Unit with 12 fiber optic cables and an MRI compatible, handheld, trackball mouse; 5) Medrad, Inc. SHS200 Power Injector; 6) InVivo Research, Inc. Precess MRI compatible patient monitor with wireless digital SPO2, ETC02, heart rate and blood pressure recording; 7) Full suite of physiological monitoring equipment from S.A. INC for small animal imaging; and 8) Microcapstar Capnograph CO2 Analyzer and MRI-1ventilator from CWE instruments for small and medium sized animals.

Computing and Data Management. The following centralized computer and file server equipment is located in the MRISC and available (1) Server, Linux, 4U Rack mounted Dell PowerEdge 6850, 64bit - 4 Quad Core Xeon Tulsa, 16GB RAM, 1.5TB SAS RAID 5 array; (2) Two Disk Array, 3U Rack mounted Dell MD1000 Power Vault, 4.5TB SAS RAID 5 array; (3) Tape Backup, 2U Rack mounted Dell TL2000, 24 x 800GB/1.6TB cartridges; (4) Network Attached Storage (NAS), 1U Rack mounted NetGear, 2.0 TB SATA RAID 5 array; (5) Dell full size 4210 rack (42U slots total; 16U slots occupied including APC; 26U slots available).

All computers and servers are protected with power supply backup and surge protecting UPSs. All MRI scans are sent to the NAS backup server immediately after the imaging session and burned to CD for permanent archiving. The MRI scanner host computer is connected to the Dell rack, containing equipment items 1-4, by 1 GB/sec fiber optic cable while the rest of the computers are connected by Cat 5e cable on a 100 MB/sec network. Institution-wide upgrades to Cat 6a network cable are currently underway. Daily incremental tape backups are made from all data on all the servers, the NAS, and the MD1000 using Yosemite Backup software running on the Poweredge 6850. Full monthly tape backups are made and stored offsite. All computers and servers are behind the UK Medical Center firewall, have individual firewalls, are accessible only with valid usernames and passwords, and have automated operating system software updating.

Bluegrass Care Clinic for HIV. The Bluegrass Care Clinic, located in Lexington, Kentucky provides HIV care, case management and psychiatric services for PLWHA in the north central Kentucky region. Currently, the clinic provides care to 1700 unique PLWHA. Approximately 175 new unique clients enroll in the clinic each year. Seventy percent of people receiving care at the Bluegrass Clinic self-report smoking cigarettes, 97% receive a prescription for anti-retroviral medication and 93% remain virally suppressed. In the Bluegrass Care Clinic there are approximately 1073 unique PLWHA, engaged in care who smoke. If we conservatively assume 1/2 may be ineligible for the study or chose not participate in the study, there are still over 500 eligible people to recruit for the study. This is nearly 2.5 times the number of people we would need to recruit (n=240) over the course of five years of the grant, if funded. These patients identify as male (81%), (18%) and transgender (1%).

The Supportive Medication Assisted Recovery Program (SMART) aims to comprehensively assess evaluation and treatment needs of patients with substance use disorders. It is housed at 245 Fountain Court and associated with the University of Kentucky. This clinic provides pharmacotherapy and psychotherapy treatment options for these patients in addition to urine drug screens and breathalyzer tests. Having 2 full time psychiatrists, 1 psychologists and 2 social workers on all days of the week, the clinic seeks to become a leader in integrative care in the state of Kentucky.

#### **Potential Risks & Benefits**

### Risks

- Describe any potential risks including physical, psychological, social, legal, ability to re-identify subjects, or other risks. Assess the seriousness and likelihood of each risk.
- Which risks may affect a subject's willingness to participate in the study?
- Describe likely adverse effects of drugs, biologics, devices or procedures participants may encounter while in the study.
- Qualitative research describe ethical issues that could arise while conducting research in the field and strategies you may use to handle those situations.
- · Describe any steps to mitigate these risks.

#### **Benefits**

- Describe potential direct benefits to study participants including diagnostic or therapeutic, physical, psychological or emotional, learning benefits. This cannot include incentives or payments.
- · State if there are no direct benefits.
- Describe potential benefits to society and/or general knowledge to be gained.

Describe why potential benefits are reasonable in relation to potential risks. If applicable, justify why risks to vulnerable subjects are reasonable to potential benefits.

The pilot study does not entail any additional risks, in addition to those already discussed for the study proper.

Study Proper. Seizure is a theoretical risk with TMS. In the Rossi et al. report it was stated that "The occurrence of seizures has been extremely rare, with most of the few new cases receiving rTMS protocols exceeding previous guidelines, often in patients under treatment with drugs which potentially lowered the seizure threshold." As Rossi et al. delineate, "rare" means that 16 cases (out of tens of thousands of rTMS sessions over the last two decades) of seizure related to rTMS have been reported. Eight occurred before safety parameters were established in 1997. Of the other eight reports, six occurred either when the safe rTMS parameters were exceeded or other safety guidelines ignored, and the actual occurrence of a seizure has been questioned in the other two (i.e., convulsive syncope or pseudoseizure may have occurred). In a workshop convened by the National Institute for Neurological Disorders and Stroke (NINDS) in 1996, researchers in the field agreed upon a set of rTMS consensus safety guidelines, including recommended stimulation parameters and contra-indications, and these consensus guidelines have been recently updated (Rossi et al., 2009). Widespread adherence to the 1996 guidelines has resulted in the virtual elimination of inadvertent seizures in rTMS studies (Rossi et al., 2009). Theta burst stimulation (TBS) that we will use in this study has been documented to be extremely safe. The risk of seizure with TBS is 0.1% (Rachid, 2017). There has been only one seizure instance reported with continuous TBS in a subject with no previous history of epilepsy but was sleep deprived after a long flight (Oberman and Pascual-Leone, 2009).

The most commonly reported side effect of rTMS is headache. This headache is typically of a muscle-tension type. It usually develops during or immediately after the stimulation and may last for minutes to hours following the end of the stimulation. It is typically limited to the day of stimulation, and usually responds promptly to single doses of over the counter pain medications. Neck pain or scalp pain may also occur. Both are usually managed easily with over-the-counter analgesics.

As noted in Rossi et al. (2009), Loo and colleagues reported mild and transient changes in auditory threshold in two depressed patients following a 2-4 week rTMS course of rTMS (16). Cases of tinnitus have been reported after rTMS treatments. In addition, recently in a study investigating the effects of rTMS on symptoms of depression, a patient experienced moderate to severe tinnitus after an rTMS session in which earplugs were not used. Rossi et al. recommended that hearing protection always should be worn during rTMS application, and that individuals with cochlear implants not receive rTMS. In the current study, earplugs will be worn by all subjects during rTMS procedures. Individuals with cochlear implants will be excluded from participation.

Risks to the unborn children of pregnant women receiving rTMS are unknown. Pregnant women will be excluded in this study. If sexually active, the subject must agree to use appropriate contraceptive measures for the duration of the study. Medically acceptable contraceptives include: (1) surgical sterilization (such as a tubal ligation or hysterectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with spermicide, or (4) an intrauterine device (IUD). Contraceptive measures such as Plan B (TM), sold for emergency use after unprotected sex, are not acceptable methods for routine use. If the subject has any uncertainty about whether they could be pregnant, another urine pregnancy test will be performed before they can participate in this protocol.

Other plausible risks include breach of confidentiality, development of suicidal thoughts and syncope (neurocardiogenic in nature). Vasodepressor (neurocardiogenic) syncope is a common reaction to anxiety and psycho-physical discomfort. It is a common experience that may occur more often than epileptic seizures during TMS testing and treatment. Suicidal thoughts have been observed to transiently develop only in subjects who have a previous history of major depressive disorder.

#### References pertinent to this section

Rossi S, Hallett M, Rossini PM, Pascual-Leone A, Safety of TMSCG. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009;120(12):2008-39. Rachid F. Safety and Efficacy of Theta-Burst Stimulation in the Treatment of Psychiatric Disorders: A Review of the Literature. J Nerv Ment Dis. 2017;205(11):823-39.

Oberman LM, Pascual-Leone A. Report of seizure induced by continuous theta burst stimulation. Brain Stimul. 2009;2(4):246-7. The pilot study will help us validate the attentional bias task to measure craving in smokers.

The study proper may benefit subjects in smoking cessation. it will also help us learn how TMS affects cognitive functions in people living with HIV who smoke. There are no known long-term health risks to the use of rTMS per se when operated within consensus safety guidelines (Rossi 2009). In 2008, the FDA approved the use of high frequency rTMS in the treatment of depression. Also in 2008, an international consensus conference on safety guidelines for rTMS (1) systematically reviewed the thousands of healthy subjects and patients who have undergone rTMS in order to allow for a better assessment of relative risks. The relative infrequency of adverse events using rTMS was noted. They concluded that in the case of Class 3 studies (studies involving indirect benefit and low risk in normal subjects and patients that are expected to yield important data on brain physiology or safety, but have no immediate relevance to clinical problems), normal volunteers should be permitted to participate in rTMS research when it is likely to produce data that are of outstanding scientific or clinical value. They also concluded that this research can be performed in a non-medical setting (i.e., psychology labs, robotics labs, research institutions, etc. as opposed to a hospital or appropriately equipped outpatient clinic). The Rossi et al. consensus report went on to suggest safety guidelines based on the now rather extensive international experience with rTMS. These guidelines include the rTMS intensity and timing parameters considered safe, training, and planning for and managing emergencies. We will follow these guidelines, and have incorporated them into our screening and session procedures.

Participation in the pilot and main parts for the study is completely voluntary, and there will be no pressure or time constraints regarding the decision to participate. If subjects experience headaches, they can withdraw without any ramifications pertaining to their respective clinic. There are no benefits to the participants except for the compensation, as well as the good will of helping the progress of scientific research. The information learned from this study may aid our understanding of the role of the TMS in modulating cognition and brain function in patients HIV and tobacco use disorder.

Rossi S, Hallett M, Rossini PM, Pascual-Leone A, Safety of TMSCG. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009;120(12):2008-39.

#### **Available Alternative Opportunities/Treatments**

Describe alternative treatments or opportunities that might be available to those who choose not to participate in the study, and which offer the subject equal or greater advantages. If applicable, this should include a discussion of the current standard of care treatment(s).

There are no alternative treatments suggested in this study

Back to Top

#### Records, Privacy, and Confidentiality

Specify where the data and/or specimens will be stored and how the researcher will ensure the privacy and confidentiality of both. Specify who will have access to the data/specimens and why they need access.

Describe how data will be managed after the study is complete:

- If data/specimens will be maintained, specify whether identifiers will be removed from the maintained information/material.
- If identifiers will not be removed, provide justification for retaining them and describe how you will protect confidentiality.
- If the data/specimens will be destroyed, verify that this will not violate <u>retention policies</u> and will adhere to applicable facility requirements.

If this study will use de-identified data from another source, describe what measures will be taken to ensure that subject identifiers are not given to the investigator.

If applicable, describe procedures for sharing data/specimens with collaborators not affiliated with UK.

For additional considerations:

Return of Research Results or Incidental Research Findings

HIPAA policies

FERPA policies

Procedures for Transfer agreements

Information regarding multi-site studies

NIH Genomic Data Sharing (GDS) Policy

Digital Data

For the pilot study, personal information collected (age, smoking history) will be will be stored in an excel sheet on a protected laptop at P336, 3rd floor, UK Department of Psychiatry at 245 Fountain Court (In a locked office and behind a protected firewall). No medical records will be reviewed for the pilot study. The excel sheets containing the personal information will be saved as an encrypted file every time, and will be stored separately from deidentified data and any other research data. Any data sharing will be restricted to the de-identified data. Data will be kept for a minimum of 7 years, and electronically destroyed by UK Policy A13-050 and UK Policy A05-055.

Study proper - Personal information of participants (Subjects' age, comorbid medical or psychiatric illnesses, history of substance use, history of traumatic brain injury/loss of consciousness, previous adverse effects with TMS, medication history, duration of treatment with suboxone, urine drug screens, breathalyzer test results) will be stored in an excel sheet on a protected laptop at P336, 3rd floor, UK Department of Psychiatry at 245 Fountain Court (In a locked office and behind a protected firewall). The excel sheets containing the personal information will be saved as an encrypted file every time. A data crosswalk of patient/participant name and MRN will be stored separately from deidentified data and any other research data. Any data sharing will be restricted to the de-identified data. Data will be kept for a minimum of 7 years, and electronically destroyed by UK Policy A13-050 and UK Policy A05-055. For the study proper, urine samples will be collected prior to every TMS session to perform drug screening.

For the pilot study, personal information of participants (age smoking history if any) will be stored in an excel sheet on a protected laptop at P336, 3rd floor, UK Department of Psychiatry at 245 Fountain Court (In a locked office and behind a protected firewall). A data crosswalk of patient/participant name and MRN will be stored separately from the deidentified data. The excel sheet containing personal information will be saved as an encrypted file every time new data is entered. Any data sharing will be restricted to the deidentified data. Data will be kept for a minimum of 7 years, and electronically destroyed by UK Policy A13-050 and UK Policy A05-055.

For the main study, personal information of participants (Age, diagnoses of seizure disorder and schizophrenia if any, history of traumatic brain injury/loss of consciousness, medication history, duration of treatment with suboxone) will be stored in an excel sheet on a protected laptop at P336, 3rd floor, UK Department of Psychiatry at 245 Fountain Court (In a locked office and behind a protected firewall). The excel sheet containing personal information will be saved as an encrypted file every time new data is entered. A data crosswalk of patient/participant name and MRN will be stored separately from the deidentified data. Any data sharing will be restricted to the de-identified data. Data will be kept for a minimum of 7 years, and electronically destroyed by UK Policy A13-050 and UK Policy A05-055. Urine samples will be collected prior to every TMS session to perform drug screening.

Before recruitment of a subject into the study we will screen the chart for seizure disorder diagnoses and schizophrenia. We will also screen for previous adverse effects to TMS. Prior to the MRI session, we will also screen for metallic implants/devices in the body. This will also be clarified with the subject.

Should a participant voice suicidal ideation at any point during the study, a thorough risk assessment would be completed immediately

and the appropriate resources would be contacted including emergency and/or outpatient resources. To mitigate CLOSE confidentiality or invasion of privacy, all procedures as part of the study will be completed at Fountain Court offices. Participant personal information and medical/psychiatric history will be stored on the University of Kentucky building at Fountain Court. Also, in order to mitigate risk of breach of confidentiality or invasion of privacy, HIPAA will be discussed with each participant at each session.

The main risks with TMS include seizures. We will screen subjects for known risk factors for seizure with rTMS (medical screening and medical history). Personnel who administer rTMS are trained to recognize a potential seizure event and to act as "first responders" to administer appropriate initial care. All study personnel will undergo basic life skills (BLS) training, and seizure-specific training. The major physical signs the study personnel will look out for in detecting a potential seizure include chewing movements, convulsions/tremor/shaking, difficulty talking, a blank stare, eyes rolling up, and profuse sweating. If any of these signs are observed, study personnel will stop the research procedure and inquire whether the subject feels okay. If the subject is unresponsive (and therefore likely experiencing a seizure), first-aid will be supplied. The first-aid response consists of making sure the subject is physically safe for the duration of the seizure. This involves moving the subjects out of the TMS chair and onto the floor lying down on his or her left side. The subject will be kept lying down on his or her left side, while the staff call emergency medical help, via a 911 call. Resources available in the laboratory include a first-aid kit and immediate phone access. A seizure constitutes a reportable adverse event, and will thus be immediately reported to the IRB via the Safety Events Form mechanism.

Initial measures for syncope are identical to those for seizures. TMS will be terminated immediately, and the subject assisted in controlled reclining without impact. Airway breathing and circulation will be assessed. Unless tonic-clonic seizure activity occurs, the subject will be turned on one side to help clear the airway and avoid aspiration.

An MRI procedure is considered to be "minimal risk" according to federal definitions. To date, no after effects have been revealed and the FDA has classified the MR procedure as possessing a "non significant risk" for the subject of study. To minimize risks, all subjects will be screened for metallic devices, implants and other contraindications to scanning. Women of child-bearing capacity will be evaluated for pregnancy using a urine pregnancy test prior to scanning. Those unlikely to tolerate the sense of confinement during scanning will also be excluded. Adequate safety monitoring and observation during scanning will be provided, as will measures to enhance the subject's physical and emotional comfort during the scan. It is possible that some subjects might experience minor distress by the confined and noisy conditions in the scanner. This possibility will be minimized by earplugs and headphones, and experienced technicians who will monitor all subjects for distress. In the event that a subject becomes anxious during a scan, the study will be halted. Subjects will be able to communicate with the investigators at all times using the intercom system should they wish to request that a study be terminated or have concerns or questions during the procedure. The subject is in full view of the operator at all times. The probability of an incidental finding that might lead to the diagnosis of an unknown abnormality is greater than zero. All subjects will be alerted to this possibility during the consent process. In that event, subjects or their designated physician will be provided copies of their anatomical scans and advised to seek further evaluation if they have concerns. Subjects will be transported between 245 Fountain Court and MRISC using UberHealth (www.uberhealth.com) operated and maintained by Department of Psychiatry.

Subjects will be transported between Fountain Court and MRISC using UberHealth. The risk associated with transportation do not exceed any risk associated with vehicle transportation in everyday life.

If subjects experience headaches they can withdraw without any ramifications pertaining to their respective clinic (Bluegrass/SMART/Beyond Birth). If subjects are hurt or get sick because of something that is done in this study, they can immediately call Gopalkumar Rakesh at 857-22-2276. After business hours, they can call the Psychiatry department On Call Group at (859) 226-7063 and explain to the physician that you are a study participant. The physician will determine what type of treatment, if any, is best for you at that time. The medical costs related to care and treatment because of research related harm will be their responsibility. The University of Kentucky Medical Center has no way to provide compensation for research subjects who receive injuries as a result of participating in biomedical and behavioral research. This means that while all investigators will do everything possible in providing careful medical care and safeguards in conducting this research, there is no way in which the institution can pay for the unlikely occurrence of injury resulting solely from the research itself.

<u>UK IRB policies</u> state that IRB-related research records must be retained for a minimum of 6 years after study closure. Do you confirm that you will retain all IRB-related records for a minimum of 6 years after study closure?

• Yes • No

Back to Top

#### **Payment**

Describe the incentives (monetary or other) being offered to subjects for their participation. If monetary compensation is offered, indicate the amount and describe the terms and schedule of payment. Please review <u>this guidance</u> for more information on payments to subjects, including restrictions and expectations.

For the pilot study, subjects would be paid \$10 for participation. Subjects will be compensated monetarily for every session of the study. For the second session of the study which could be TBS or sham TMS, they will receive \$120 and for the third session of the study which could be active or sham, they will receive \$150.

#### Costs to Subjects
Include a list of services and/or tests that will not be paid for by the sponsor and/or the study (e.g., MRI, HIV). Keek subject will not know what is "standard" – and thus not covered by the sponsor/study – unless you tell them.

There will be no cost to the subject to participate in the pilot or main research studies.

## **Data and Safety Monitoring**

The IRB requires review and approval of data and safety monitoring plans for greater than minimal risk research or NIH-funded/FDA-regulated clinical investigations.

- If you are conducting greater than minimal risk research, or your clinical investigation is NIH-funded, describe your Data and Safety Monitoring Plan (DSMP). Click here for additional guidance on developing a Data and Safety Monitoring Plan.
- If this is a non-sponsored investigator-initiated protocol considered greater than minimal risk research, and if you are planning on using a Data and Safety Monitoring Board (DSMB) as part of your DSMP, <u>click here for additional guidance</u> for information to include with your IRB application.



For both the pilot study and the study proper, subject data will be de-identified and stored on a spreadsheet on the computer in Fountain Court P336 in a locked office and behind a firewall. The excel sheet containing the personal information will be saved as an encrypted file every time. A data crosswalk of patient/participant name and MRN will be stored separately from deidentified data and any other research data. Prior to administering TMS, all personnel will be trained with the machine. The PI has been trained in TMS from Duke University Medical Center, NC. One of the other co-investigators on the study, Michael Wesley has a TMS suite and will collaborate with the PI to set up safety monitoring and adverse event reporting policies. In addition the PI will work closely with consultants from Duke/NIMH and the research officer with TMS manufacturer Magventure to administer safety monitoring policies for this study. We will institute procedures for promptly detecting harm and mitigating potential injuries. This will also ensure adequate feedback of information to all investigators. Any data sharing will be restricted to the de-identified data. Data will be kept for a minimum of 7 years, and electronically destroyed by UK Policy A13-050 and UK Policy A05-055.

Any adverse events or unanticipated problems would be reported per the IRB's policy on "Unanticipated Problem and Safety Reporting." https://www.research.uky.edu/uploads/ori-d20000-irb-policy-unanticipated-problem-and-safety-reporting-pdf

# Future Use and Sharing of Research Data

If the results of this study will be used by members of the research team or shared with other researchers for future studies, please address the following:

- list the biological specimens and/or information that will be kept
- briefly describe the types, categories and/or purposes of the future research
- describe any risks of the additional use
- describe privacy/confidentiality protections that will be put into place
- describe the period of time specimens/information may be used
- · describe procedures for sharing specimens/information with secondary researchers
- describe the process for, and limitations to, withdrawal of specimens/data

## WILL YOUR INFORMATION (OR SPECIMEN SAMPLES) BE USED FOR FUTURE RESEARCH?

All identifiable information (e.g., your name, medical record number, or date of birth) will be removed from the information or samples collected in this study. This means that no link or code to your identity will be kept. After all identifiers have been removed, the information or samples may be used for future research or shared with other researchers without your additional informed consent, Once you give your permission to have your deidentified information or samples stored, they will be available indefinitely and cannot be removed due to the inability to identify them.

#### AUTHORIZATION TO USE OR DISCLOSE YOUR IDENTIFIABLE HEALTH INFORMATION

The privacy law, HIPAA (Health Insurance Portability and Accountability Act), requires researchers to protect your health information. The following sections of the form describe how researchers may use your health information. Your health information that may be accessed, used and/or released includes:

Age, diagnoses of seizure disorder and schizophrenia if any, history of traumatic brain injury/loss of consciousness, medication history, duration of treatment with suboxone. The diagnoses in your chart will be looked at since these form part of inclusion criteria for the study. We would like to know how long you have been on suboxone as that would be used as a predictor variable in analyses of results from the study.

The Researchers may use and share your health information with:

- The University of Kentucky's Institutional Review Board/Office of Research Integrity;
- · Law enforcement agencies when required by law;
- University of Kentucky representatives;
- UK Hospital
- Food and Drug Administration

The researchers agree to only share your health information with the people listed in this document. Should your health information be released to anyone that is not regulated by the privacy law, your health information may be

shared with others without your permission; however, the use of your health information may still be regulated by applicable federal and state laws.

You may not be allowed to participate in the research study if you do not sign this form. If you decide not to sign this form, it will not affect your:

Current or future healthcare at the University of Kentucky;

Current or future payments to the University of Kentucky;

- · Ability to enroll in any health plans (if applicable); or
- Eligibility for benefits (if applicable).

Are you recruiting or expect to enroll **Non-English Speaking Subjects or Subjects from a Foreign Culture**? (does not include short form use for incidentally encountered non-English subjects)

• Yes • No

Non-English Speaking Subjects or Subjects from a Foreign Culture

#### **Recruitment and Consent:**

Describe how information about the study will be communicated to potential subjects appropriate for their culture, and if necessary, how new information about the research may be relayed to subjects during the study.

When recruiting Non-English-speaking subjects, provide a consent document in the subject's primary language. After saving this section, attach both the English and translated consent documents in the "Informed Consent" section.

## **Cultural and Language Consultants:**

The PI is required to identify someone who is willing to serve as the cultural consultant to the IRB.

- This person should be familiar with the culture of the subject population and/or be able to verify that translated documents are the equivalent of the English version of documents submitted.
- The consultant should not be involved with the study or have any interest in its IRB approval.
- Please include the name, address, telephone number, and email of the person who agrees to be the cultural consultant for your study.
- ORI staff will facilitate the review process with your consultant. Please do not ask them to review your protocol separately.

For more details, see the IRB Application Instructions on Research Involving Non-English Speaking Subjects or Subjects from a Foreign Culture.

## Local Requirements:

If you will conduct research at an international location, identify and describe:

- relevant local regulations
- · data privacy regulations
- · applicable laws
- ethics review requirements for human subject protection

Please provide links or sources where possible. If the project has been or will be reviewed by a local ethics review board, attach a copy in the "Additional Information/Materials" section. You may also consult the current edition of the <a href="International Compilation of Human Research Standards">International Compilation of Human Research Standards</a>

Does your study involve HIV/AIDS research and/or screening for other reportable diseases (e.g., Hepatitis C, etc...)?

⊙ Yes ○ No

HIV/AIDS Research

If you have questions about what constitutes a reportable disease and/or condition in the state of Kentucky, see ORI's summary sheet: "Reporting Requirements for Diseases and Conditions in Kentucky" [PDF].

**HIV/AIDS Research:** There are additional IRB requirements for designing and implementing the research and for obtaining informed consent. Describe additional safeguards to minimize risk to subjects in the space provided below.

For additional information, visit the online <u>IRB Survival Handbook</u> to download a copy of the "Medical IRB's requirements for Protection of Human Subjects in Research Involving HIV Testing" [D65.0000] <u>[PDF]</u>, and visit the <u>Office for Human Research Protections web site</u> for statements on AIDS research, or contact the Office of Research Integrity at 859-257-9428.

Although the research project involves subjects with a diagnosis of HIV/AIDS, we will not perform HIV testing in these subjects.

#### PI-Sponsored FDA-Regulated Research

Is this an investigator-initiated study that:

Back to Top

- 1) involves testing a Nonsignificant Risk (NSR) Device, or
- 2) is being conducted under an investigator-held Investigational New Drug (IND) or Investigational Device Exemption (IDE)?

PI-Sponsored FDA-Regulated Research

If the answer above is yes, then the investigator assumes the regulatory responsibilities of both the investigator and sponsor. The Office of Research Integrity provides a summary list of sponsor IND regulatory requirements for drug trials [PDF], IDE regulatory requirements for SR device trials [PDF], and abbreviated regulatory requirements for NSR device trials [PDF]. For detailed descriptions see FDA Responsibilities for Device Study Sponsors or FDA Responsibilities for IND Drug Study Sponsor-Investigators.

- Describe the experience/knowledge/training (if any) of the investigator serving as a sponsor (e.g., previously held an IND/IDE); and
- Indicate if any sponsor obligations have been transferred to a commercial sponsor, contract research organization (CRO), contract monitor, or other entity (provide details or attach FDA 1571).

One of the other co-investigators on the study, Michael Wesley has a TMS suite and will collaborate with the PI to set up safety monitoring and adverse event reporting policies. In addition the PI will work closely with consultants from Duke/NIMH and the research officer with TMS manufacturer Magventure to administer safety monitoring policies for this study. The PI has received TMS training from Duke University, NC. The PI has also taken required CITI courses needed for the role, which are attached herewith.

In accordance with FDA requirements for investigators who are sponsors of non significant risk devices, the PI will label the TMS device with the statement "CAUTION - Investigational Device. Limited by Federal (or United States) law to investigational use." (21 CFR 812.5). The PI will obtain IRB approval before using the device and will maintain IRB approval for the device during its period of use. The PI will also ensure that investigator(s) are complying with FDA, IRB and sponsor requirements. (21 CFR 812.46). The PI will conduct an evaluation of unanticipated adverse events and terminate the study if necessary. (21 CFR 812.46). The PI will resume terminated studies only after receiving approval from the IRB and if terminated due to an unanticipated adverse device effect, also obtain FDA approval to resume the study. (21 CFR 812.46). The PI will ensure that each investigator obtains consent for each subject unless the IRB grants a waiver under 21 CFR 56.109(c). The PI will also ensure that each investigator maintains accurate and complete records in accordance with FDA regulations and reports the results to the appropriate parties. (21 CFR 812.140 & 21 CFR 812.150). The PI will permit and facilitate monitoring and auditing by the IRB or inspection by federal or state regulatory agencies as appropriate. (21 CFR 812.145). The PI will limit promotion of the device and register the study at ClinicalTrials.gov per the Food and Drug Administration Amendments Act (FDAAA) of 2007 (Public Law 110-85). The PI will also comply with FDA reg

IRB policy requires mandatory training for all investigators who are also FDA-regulated sponsors (see <u>Sponsor-Investigator FAQs</u>). A sponsor-investigator must complete the applicable Office of Research Integrity web based training, (drug or device) before final IRB approval is granted.

If the sponsor-investigator has completed equivalent sponsor-investigator training, submit documentation of temporary larger training and the submit documentation of temporary larger training and the submit documentation of the submit documentation of the submit documentation of the submit documentation and the submit documentation of the submit documentation and the submit docume

# Attachments

| Attach Type | File Name |
|--------------------|-------------------------------------|
| SponsorInvTraining | 62379_SponsorInvTraining_266756.pdf |
| SponsorInvTraining | 62379_SponsorInvTraining_266757.pdf |
| SponsorInvTraining | 62379_SponsorInvTraining_266758.pdf |
| SponsorInvTraining | 62379_SponsorInvTraining_266759.pdf |
| SponsorInvTraining | 62379_SponsorInvTraining_266760.pdf |
| SponsorInvTraining | 62379_SponsorInvTraining_266763.pdf |
| SponsorInvTraining | 62379_SponsorInvTraining_266763.pdf |

HIPAA 0 unresolved comment(s)

(Visit ORI's <u>Health Insurance Portability and Accountability Act (HIPAA) web page</u> to determine if your research falls under the HIPAA Privacy Regulation.)

If yes, check below all that apply and attach the applicable document(s):

☐ HIPAA De-identification Certification Form 

✓ HIPAA Waiver of Authorization

Attachments

| Attach Type | File Name |
|-------------|-------------------------------------------------------|
| Waiver | ori-f10700-form-k-hipaa-waiver-authorization-word.pdf |

# STUDY DRUG INFORMATION

0 unresolved comment(s)

## The term drug may include:

- FDA approved drugs,
- unapproved use of approved drugs,
- investigational drugs or biologics,
- other compounds or products intended to affect structure or function of the body, and/or
- <u>complementary and alternative medicine products</u> such as dietary supplements, substances generally recognized as safe (GRAS) when used to diagnose, cure mitigate, treat or prevent disease, or clinical studies of <u>e-cigarettes</u> examining a potential therapeutic purpose.

Does this protocol involve a drug including an FDA approved drug; unapproved use of an FDA approved drug; and/or an investigational drug?

Yes 
 No

If yes, complete the questions below. Additional study drug guidance.

| Drug Name: | |
|---|---|
| Oncology or Non-Oncology). | quired by Hospital Policy to utilize <u>Investigational Drug Service (IDS) pharmacies</u> . Use of IDS is highly recommended, but optional for outpatient studies. Outpatient is are subject to periodic inspection by the IDS for compliance with drug accountability |
| ndicate where study drug(s) | will be housed and managed: |
| Investigational Drug Se | ervice (IDS) UK Hospital |
| Other Location: | |
| Is the study being conducted | under a valid Investigational New Drug (IND) application? |
| CYes CNo | |
| If Yes, list IND #(s) and | complete the following: |
| 11 100, 1101 1112 11(0) dilid | osimplete the following. |
| IND Submitted/Held by: | |
| IND Submitted/Held by:<br>Sponsor: □ | Held By: |
| · | |
| Sponsor: □ | Held By: |
| Sponsor: □ Investigator: □ | Held By: |
| Sponsor: Investigator: Other: Checkmark if the stu | Held By: |
| Sponsor: Investigator: Other: Checkmark if the stu | Held By: Held By: Held By: Held By: dy is being conducted under FDA's Expanded Access Program (e.g., Treatment |
| Sponsor: Investigator: Other: Checkmark if the stu IND) or if this is an Indi FDA's Expanded Acce attach the following: FDA Form 3926; FDA expanded acce | Held By: Held By: Held By: dy is being conducted under FDA's Expanded Access Program (e.g., Treatment vidual Patient Expanded Access IND (FDA Form 3926). |

Complete and attach the required <u>Study Drug Form</u> picking "Study Drug Form" for the document type. Any applicable drug documentation (e.g., Investigator Brochure; approved labeling; publication; FDA correspondence, etc.) should be attached using "Other Drug Documentation" for the document type.



Attachments

## STUDY DEVICE INFORMATION

0 unresolved comment(s)

## A DEVICE may be a:

- · component, part, accessory;
- · assay, reagent, or in-vitro diagnostic device;
- software, digital health, or mobile medical app;
- other instrument if intended to affect the structure or function of the body, diagnose, cure, mitigate, treat or prevent disease; or
- a homemade device developed by an investigator or other non-commercial entity and not approved for marketing by FDA.

For additional information, helpful resources, and definitions, see ORI's <u>Use of Any Device Being Tested in Research web page</u>.

Does this protocol involve testing (collecting safety or efficacy data) of a medical device including an FDA approved device, unapproved use of an approved device, humanitarian use device, and/or an investigational device?

Yes ○ No

[Note: If a marketed device(s) is only being used to elicit or measure a physiologic response or clinical outcome, AND, NO data will be collected on or about the device itself, you may answer "no" above, save and exit this section, (Examples: a chemo drug study uses an MRI to measure tumor growth but does NOT assess how effective the MRI is at making the measurement; an exercise study uses a heart monitor to measure athletic performance but no safety or efficacy information will be collected about the device itself, nor will the data collected be used for comparative purposes against any other similar device).]

If you answered yes above, please complete the following questions.

| 0 | th | ei | •• | F |
|---|----|----|----|---|

Held By: NA

 $\Box$  Check if this is a Treatment IDE or Compassionate Use under the Food and Drug Administration (FDA) Expanded Access program.

For Individual or Small Group Expanded Access, see <u>FDA's Early Expanded Access Program Information</u>, and attach the following:

- FDA expanded access approval or sponsor's authorization;
- An independent assessment from an uninvolved physician, if available;
- Confirmation of agreement from manufacturer or entity authorized to provide access to the product.

For guidance and reporting requirements at the conclusion of treatment see the Medical Device SOP.

Does the intended use of any research device being tested (not clinically observed) in this study meet the regulatory <u>definition</u> of Significant Risk (SR) device?

- c Yes. Device(s) as used in this study presents a potential for serious risk to the health, safety, or welfare of a subject and (1) is intended as an implant; or (2) is used in supporting or sustaining human life; or (3) is of substantial importance in diagnosing, curing, mitigating or treating disease, or otherwise prevents impairment of human health; or (4) otherwise presents a potential for serious risk to the health, safety, or welfare of a subject.

Complete and attach the required <u>Study Device Form</u>, picking the "Study Device Form" for the document type. Any applicable device documentation (e.g., Manufacturer information; patient information packet; approved labeling; FDA correspondence, etc.) should be attached using "Other Device Documentation" for the document type.



# Attachments

| Attach Type | File Name |
|-------------------|--------------------|
| Study Device Form | MagVentureX100.pdf |
| Study Device Form | IRB IDE device.pdf |

## RESEARCH SITES

0 unresolved comment(s)

To complete this section, ensure the responses are accurate then click "SAVE".

A) Check all the applicable sites listed below at which the research will be conducted. If none apply, you do not need to check any boxes.

#### **UK Sites**

- □ UK Classroom(s)/Lab(s)
- UK Clinics in Lexington
- □ UK Clinics outside of Lexington
- □ UK Healthcare Good Samaritan Hospital
- □ UK Hospital

#### -Schools/Education Institutions

- □ Fayette Co. School Systems \*
- ☐ Other State/Regional School Systems
- □ Institutions of Higher Education (other than UK)

\*Fayette Co. School systems, as well as other non-UK sites, have additional requirements that must be addressed. See ORI's <u>IRB Application Instructions</u> - <u>Off-site Research</u> web page for details.

## Other Medical Facilities

- □ Bluegrass Regional Mental Health Retardation Board
- ☐ Cardinal Hill Hospital
- □ Eastern State Hospital
- □ Norton Healthcare
- □ Nursing Homes
- □ Shriner's Children's Hospital
- □ Veterans Affairs Medical Center
- □ Other Hospitals and Med. Centers
- □ Correctional Facilities
- ☐ Home Health Agencies
- □ International Sites

Research activities conducted at performance sites that are not owned or operated by the University of Kentucky, at sites that are geographically separate from UK, or at sites that do not fall under the UK IRB's authority, are subject to special procedures for coordination of research review. Additional information is required (see IRB Application Instructions - Off-Site Research web page), including:

- A letter of support and local context is required from non-UK sites. See Letters of Support and Local Context on the IRB Application Instructions Off-Site Research web page for more information.
- Supportive documentation, including letters of support, can be attached below.
- NOTE: If the non-UK sites or non-UK personnel are engaged in the research, there are additional federal and university requirements which need to be completed for their participation. For instance, the other site(s) may need to complete their own IRB review, or a cooperative review arrangement may need to be established with non-UK

| _ | :1 |
|---|------|
| • | ITAC |

Questions about the participation of non-UK sites/personnel should be discussed with the ORI staff at (859) 257-9428.

| List all other r | on-UK owned/operated | locations where th | e research will be o | conducted: | |
|---|---|---|---|---|---|
| Describe the | role of any non-UK site(s | s) or non-UK perso | nne <b>l</b> who will be pa | rticipating in your rese | earch. |
| Attachments | | | | | |
| ls this a multi-site s | tudy for which <b>you are</b> | the lead investiga | itor or UK is the l | ead site? ⊜Yes ଜ No | ı |
| | e plan for the managementerim results from the n | | anticipated prob <b>l</b> en | ns, noncomp <b>l</b> iance, ar | nd submission of protoco |

C) If your research involves collaboration with any sites and/or personnel outside the University of Kentucky, then it is considered multisite research and IRB reliance issues will need to be addressed. This may include national multi-center trials as well local studies involving sites/personnel external to UK. If you would like to request that the University of Kentucky IRB (UK IRB) serve as the lead IRB for your study, or if you would like the UK IRB to defer review to another IRB, please contact the <a href="mailto:IRBReliance@uky.edu">IRBReliance@uky.edu</a>.

## **RESEARCH ATTRIBUTES**

0 unresolved comment(s)

Indicate the items below that apply to your research. Depending on the items applicable to your research, you may be required to complete additional forms or meet additional requirements. Contact the ORI (859-257-9428) if you have questions about additional requirements.

□ Not applicable

# -Check All That Apply-

- □ Academic Degree/Required Research
- □ Alcohol/Drug/Substance Abuse Research
- □ Biological Specimen Bank Creation (for sharing)
- ☐ Cancer Research
- CCTS-Center for Clinical & Translational Science
- □ Certificate of Confidentiality
- □ Clinical Research
- □ Clinical Trial Phase 1
- Clinical Trial
- □ Collection of Biological Specimens for internal banking and use (not sharing)
- □ Community-Based Participatory Research
- □ Deception
- □ Educational/Student Records (e.g., GPA, test scores)
- ☐ Emergency Use (Single Patient)
- ☐ Gene Transfer
- ☐ Genetic Research
- $\sqcap$  GWAS (Genome-Wide Association Study) or NIH Genomic Data Sharing (GDS)
- □ Human Cells, Tissues, and Cellular and Tissue Based Products
- □ Individual Expanded Access or Compassionate Use
- □ International Research
- □ Planned Emergency Research Involving Exception from Informed Consent
- □ Recombinant DNA
- □ Registry or data repository creation
- ☐ Stem Cell Research
- □ Suicide Ideation or Behavior Research
- ☐ Survey Research
- □ Transplants
- $\hfill\Box$  Use, storage and disposal of radioactive material and radiation producing devices
- □ Vaccine Trials

For additional requirements and information:

- Cancer Research (MCC PRMC)
- <u>Certificate of Confidentiality</u> (look up "Confidentiality/Privacy...")
- <u>CCTS (Center for Clinical and Translational</u> Science)
- <u>Clinical Research</u> (look up "What is the definition of....)
- Clinical Trial
- Collection of Biological Specimens for Banking (look up "Specimen/Tissue Collection...")
- <u>Collection of Biological Specimens</u> (look up "Specimen/Tissue Collection...")
- Community-Based Participatory Research (look up "Community-Engaged...")
- Data & Safety Monitoring Board (DSMB)

\*For Medical IRB: <u>Service Request Form</u> for CCTS DSMB

- Data & Safety Monitoring Plan
- Deception\*

\*For deception research, also go to the E-IRB Application Informed Consent section, checkmark and complete "Request for Waiver of Informed Consent Process"

- Emergency Use (Single Patient) [attach Emergency Use Checklist] (PDF)
- Genetic Research (look up "Specimen/Tissue Collection...")
- Gene Transfer
- <u>HIV/AIDS Research</u> (look up "Reportable Diseases/Conditions")
- Screening for Reportable Diseases [E2.0000] (PDF)
- International Research (look up "International & Non-English Speaking")
- NIH Genomic Data Sharing (GDS) Policy (PDF)
- Planned Emergency Research Involving Waiver of Informed Consent\*

\*For Planned Emergency Research Involving Waiver of Informed Consent, also go to the E-IRB Application Informed Consent section, checkmark and complete "Request for Waiver of Informed Consent Process"

• <u>Use, storage and disposal of radioactive material</u> and radiation producing devices

# **FUNDING/SUPPORT**

0 unresolved comment(s)

If the research is being submitted to, supported by, or conducted in cooperation with an external or internal agency or funding program, indicate below all the categories that apply. ①

□ Not applicable

| Check All That Apply——————————————————————————————————— | |
|---|---|
| ☐ Grant application pending | Click applicable listing(s) for additional requirements and information: |
| ☐ (HHS) Dept. of Health & Human Services | Click applicable listing(s) for additional requirements and information. |
| □ (NIH) National Institutes of Health | (HHS) Dept. of Health & Human Services |
| ` , | (NIH) National Institutes of Health |
| | (CDC) Centers for Disease Control & Prevention (HRSA) Health Resources & Services Administration |
| ☐ (HRSA) Health Resources and Services | (SAMHSA) Substance Abuse & Mental Health Services |
| Administration | Administration |
| □ (SAMHSA) Substance Abuse and Mental | Industry (Other than Pharmaceutical Companies) [IRB Fee Info] |
| Health Services Administration | <u>National Science Foundation</u> |
| □(DoJ) Department of Justice or Bureau of | <ul> <li>(DoEd) U.S. Department of Education</li> </ul> |
| Prisons | (DoJ) Department of Justice or Bureau of Prisons |
| □(DoE) Department of Energy | (DoE) Department of Energy Summary and Department of Energy<br>Identifiable Information Compliance Checklist |
| □(EPA) Environmental Protection Agency | (EPA) Environmental Protection Agency |
| □ Federal Agencies Other Than Those Listed | 1 (ELT 71) ETIVILOTITION ATT TOLOGISTI / I GOTTO Y |
| Here | |
| □ Industry (Other than Pharmaceutical | |
| Companies) | |
| Internal Grant Program w/ proposal | |
| □ Internal Grant Program w/o proposal | |
| □ National Science Foundation | |
| □ Other Institutions of Higher Education | |
| □ Pharmaceutical Company | |
| □ Private Foundation/Association | |
| □U.S. Department of Education | |
| □State | |
| Other: | |
| Specify the funding source and/or cooperating | organization(s) (e.g., National Cancer Institute, Ford Foundation, Eli Lilly |
| & Company, South Western Oncology Group, E | |
| NA | |

## -Add Related Grants-

If applicable, please search for and select the OSPA Account number or Electronic Internal Approval Form (eIAF) # (notif #) associated with this IRB application using the "Add Related Grants" button.

If required by your funding agency, upload your grant using the "Grant/Contract Attachments" button.

Add Related Grants

**Grant/Contract Attachments** 

The research involves use of Department of Defense (DoD) funding, military personnel, DoD facilities, or other (See <u>DoD SOP</u> and <u>DoD Summary</u> for details)

Yes 
 No

Using the "attachments" button (below), attach applicable materials addressing the specific processes described in the DoD SOP.

**DOD SOP Attachments** 

Additional Certification: (If your project is federally funded, your funding agency may request an Assurance/ Certification/Declaration of Exemption form.) Check the following if needed:

□ Protection of Human Subjects Assurance/Certification/Declaration of Exemption (Formerly Optional Form – 310)

Assurance/Certification Attachments

## **OTHER REVIEW COMMITTEES**

0 unresolved comment(s)

If you check any of the below committees, additional materials may be required with your application submission.

Does your research fall under the purview of any of the other review committees listed below? [If yes, check all that apply and attach applicable materials using the attachment button at the bottom of your screen.]

Yes No

#### **Additional Information**

- □ Institutional Biosafety Committee
- □ Radiation Safety Committee
- □ Radioactive Drug Research Committee
- ☐ Markey Cancer Center (MCC) Protocol Review and Monitoring Committee (PRMC)
- ☐ Graduate Medical Education Committee (GME)
- ☐ Office of Medical Education (OME)
- Institutional Biosafety Committee (IBC) Attach required IBC materials
- Radiation Safety Committee (RSC) For applicability, see instructions and attach form
- Radioactive Drug Research Committee (RDRC)
- Markey Cancer Center (MCC) Protocol Review and Monitoring <u>Committee (PRMC)\*\*</u> - Attach MCC PRMC materials, if any, per instructions.
- Office of Medical Education (OME)
- Graduate Medical Education Committee (GME)

# Attachments

\*\* If your study involves cancer research, be sure to select "Cancer Research" in the "Research Attributes" section. ORI will send your research protocol to the Markey Cancer Center (MCC) Protocol Review and Monitoring Committee (PRMC). The MCC PRMC is responsible for determining whether the study meets the National Cancer Institute (NCI) definition of a clinical trial and for issuing documentation to you (the investigator) which confirms either that PRMC approval has been obtained or that PRMC review is not required. Your IRB application will be processed and reviewed independently from the PRMC review.

## ADDITIONAL INFORMATION/MATERIALS

0 unresolved comment(s)

Do you want specific information inserted into your approval letter? O Yes @ No

Approval Letter Details:

If you wish to have specific language included in your approval letter (e.g., serial #, internal tracking identifier, etc...), type that language in the box below exactly as it should appear in the letter. The text you enter will automatically appear at the top of all approval letters, identical to how you typed it, until you update it. Don't include instructions or questions to ORI staff as those will appear in your approval letter. If these details need to be changed for any reason, you are responsible for updating the content of this field.

| Additions | al N/ | اعtد | ria | e. |
|-----------|-------|------|-----|----|

If you have other materials you would like to include for the IRB's consideration, check all that apply and attach the corresponding documents using the Attachments button below.

- □ Detailed protocol
- □ Dept. of Health & Human Services (DHHS) approved protocol (such as NIH sponsored Cooperative Group Clinical Trial)
- ☐ Other Documents

## Protocol/Other Attachments

| Attach Type File Name | |
|---|---|
| Protocol | CC-OD-21-1789.pdf |
| Protocol | RE_IRB# 64473 TMS for Smoking Cessation in PLWHA.pdf |

NOTE: Instructions for Dept. of Health & Human Services (DHHS)-approved protocol

If you have password protected documents, that feature should be disabled prior to uploading to ensure access for IRB review.

To view the materials currently attached to your application, click "All Attachments" on the left menu bar.

## **SIGNATURES (ASSURANCES)**

0 unresolved comment(s)

All IRB applications require additional assurances by a Department Chairperson or equivalent (DA), and when applicable, a Faculty Advisor or equivalent (FA). This signifies the acceptance of certain responsibilities and that the science is meritorious and deserving of conduct in humans. The person assigned as DA should not also be listed in the Study Personnel section, and the individual assigned as FA should be listed in the Study Personnel section.

For a list of responsibilities reflected by signing the Assurance Statement, refer to "What does the Department Chairperson's Assurance Statement on the IRB application mean?"

# **Required Signatures:**

| 0 | | | | | |
|---|---|---|---|---|---|
| First Name | Last<br>Name | Role | Department | Date<br>Signed | |
| Seth | Himelhoch | Department<br>Authorization | Psychiatry | 02/10/2021<br>08:09 AM | View/Sign |
| Gopalkumar | Rakesh | Principal<br>Investigator | Psychiatry | 02/08/2021<br>05:06 PM | View/Sign |

#### Department Authorization

▼ This is to certify that I have reviewed this research protocol and that I attest to the scientific validity and importance of this study; to the qualifications of the investigator(s) to conduct the project and their time available for the project; that facilities, equipment, and personnel are adequate to conduct the research; and that continued guidance will be provided as appropriate. When the principal investigator assumes a sponsor function, the investigator has been notified of the additional regulatory requirements of the sponsor and by signing the principal investigator Assurance Statement, confirms he/she can comply with them.

\*If the Principal Investigator is also the Chairperson of the department, the Vice Chairperson or equivalent should complete the "Department Authorization".

\*\*IF APPLICABLE FOR RELIANCE: I attest that the principal investigator has been notified of the regulatory requirements of both the Reviewing and Relying IRBs, according to the information provided in the E-IRB application. The attached Reliance Assurance Statement, signed by the principal investigator, confirms that he/she can comply with both sets of IRB requirements.

-Principal Investigator's Assurance Statement

I understand the University of Kentucky's policies concerning research involving human subjects and I agree:

- 1. To comply with all IRB policies, decisions, conditions, and requirements;
- 2. To accept responsibility for the scientific and ethical conduct of this research study;
- 3. To obtain prior approval from the Institutional Review Board before amending or altering the research protocol or implementing changes in the approved consent/assent form;
- 4. To report to the IRB in accord with IRB/IBC policy, any adverse event(s) and/or unanticipated problem(s) involving risks to subjects;
- 5. To complete, on request by the IRB for Full and Expedited studies, the Continuation/Final Review Forms;
- 6. To notify the Office of Sponsored Projects Administration (OSPA) and/or the IRB (when applicable) of the development of any financial interest not already disclosed:
- 7. Each individual listed as study personnel in this application has received the mandatory human research protections education (e.g., CITI);
- 8. Each individual listed as study personnel in this application possesses the necessary experience for conducting research activities in the role described for this research study.
- 9. To recognize and accept additional regulatory responsibilities if serving as both a sponsor and investigator for FDA regulated research.

- I have appropriate facilities and resources for conducting the study;
- I am aware of and take full responsibility for the accuracy of all materials submitted to the IRB for review;
- If applying for an exemption, I also certify that the only involvement of human subjects in this research study will be in the categories specified in the Protocol Type: Exemption Categories section.
- If applying for an Abbreviated Application (AA) to rely on an external IRB, I understand that certain items above (1, 3, 4, 7-8) may not apply, or may be altered due to external institutional/IRB policies. I document my agreement with the <a href="Principal Investigator Reliance Assurance Statement">Principal Investigator Reliance Assurance Statement</a> by digitally signing this application.

\*You will be able to "sign" your assurance after you have sent your application for signatures (use Submission section). Please notify the personnel required for signing your IRB application after sending for signatures. Once all signatures have been recorded, you will need to return to this section to submit your application to ORI.

## **SUBMISSION INFORMATION**

0 unresolved comment(s)

\*\*\* If this Continuation Review entails a change in the scope of your activities to include COVID-19 related research, please insert "COVID19" at the start of your Project and Short Titles.\*\*\*

Each Section/Subsection in the menu on the left must have a checkmark beside it (except this Submission section) indicating the Section/Subsection has been completed. Otherwise your submission for IRB review and approval cannot be sent to the Office of Research Integrity/IRB.

If applicable, remember to update the Approval Letter Details text box under the Additional Information section

If your materials require review at a convened IRB meeting which you will be asked to attend, it will be scheduled on the next available agenda and you will receive a message to notify you of the date.

If you are making a change to an attachment, you need to delete the attachment, upload a highlighted version that contains the changes (use Document Type of "Highlighted Changes"), and a version that contains the changes without any highlights (use the appropriate Document Type for the item(s)). Do **not** delete approved attachments that are still in use.

-Principal Investigator's Assurance Statement-

I understand the University of Kentucky's policies concerning research involving human subjects, and I attest to:

- 1. Having reviewed all the investigational data from this study, including a compilation of all internal and external unanticipated problems.
- 2. Having reviewed, if applicable, information from the sponsor including updated investigator brochures and data and safety monitoring board reports.

I also attest that I have reviewed pertinent materials concerning the research and concluded:

• The human subject risk/benefit relationship is unaffected, mitigated, or eliminated by closure of the study and all pertinent materials for closure of the research are being submitted to the IRB for consideration.

■ By checking this box, I am providing assurances for the applicable items listed above.

Your protocol has been submitted.





# Consent and Authorization to Participate in a Research Study

**KEY INFORMATION FOR** Transcranial Magnetic Stimulation (TMS) for Smoking Cessation for People Living with HIV/AIDS (PLWHA)

We are asking you to choose whether or not to volunteer for a research study about the effects of non-invasive, non-significant risk transcranial magnetic stimulation on how your brain makes decisions and focusses attention. We are asking you because you fulfill eligibility criteria for the study. You are also being asked to participate because you have expressed interest in participating in this study, and because you passed the medical screen. If you volunteer to take part in this study, you will be one of about 30 people to do so at the University of Kentucky. This page is to give you key information to help you decide whether to participate. We have included detailed information after this page. Ask the research team questions. If you have questions later, the contact information for the research investigator in charge of the study is below.

# WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST?

The purpose of this study is to learn more about how non-invasive, non-significant risk transcranial magnetic stimulation influences the brain's decision-making process and visual attention in people living with HIV. By doing this study, we hope to learn how the brain chooses short term versus long term rewards, in addition to learning how your eyes focus attention when seeing images related to smoking versus neutral images. Your participation in this research will last about three days. This is a research project, not a treatment program. The transcranial stimulation we use is called transcranial magnetic stimulation (TMS). In this study, TMS will be used in a manner which is an investigational procedure, aimed at temporarily changing the way that a part of your brain works. TMS has been approved by the Food and Drug Administration (FDA) as a treatment for depression, but in this study TMS is being used to investigate if changes in the activities of certain areas of the brain affect memory. Although the form of TMS we use has not been approved by FDA for smoking cessation, another type of TMS called deep TMS has been approved by the FDA. You will also be asked to undergo brain MRI scans before and after the TMS session.

## WHAT ARE KEY REASONS YOU MIGHT CHOOSE TO VOLUNTEER FOR THIS STUDY?

This research study may have direct benefit to you for smoking cessation. The study will inform us about how transcranial magnetic stimulation affects cognitive functions in tobacco use. For a complete description of benefits, refer to the Detailed Consent.

# WHAT ARE KEY REASONS YOU MIGHT CHOOSE NOT TO VOLUNTEER FOR THIS STUDY?

This study requires you to come to 245 Fountain Court for one day and to Magnetic Resonance Imaging and Spectroscopy Center (MRISC) for one day. If this will be an issue, you may not want to volunteer for this study. For a complete description of risks from the study, refer to the Detailed Consent and/or Appendix. If you experience headaches from the TMS procedure, you can withdraw from the study without ramifications regarding your clinical care.

## DO YOU HAVE TO TAKE PART IN THE STUDY?

If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits or rights you would normally have if you choose not to volunteer.

# WHAT IF YOU HAVE QUESTIONS, SUGGESTIONS OR CONCERNS?

If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study contact Gopalkumar Rakesh MD, Assistant Professor, Department of Psychiatry at 857-222-2276 during regular business hours. If outside regular business hours, please contact the Psychiatry department On Call Group at (859) 226-7063 and explain to the physician that you are a study participant.

If you have any concerns or questions about your rights as a volunteer in this research, contact staff in the University of Kentucky (UK) Office of Research Integrity (ORI) between the business hours of 8am and 5pm EST, Monday-Friday at 859-257-9428 or toll free at 1-866-400-9428.

## **DETAILED CONSENT:**

# ARE THERE REASONS WHY YOU WOULD NOT QUALIFY FOR THIS STUDY?

You should not participate if you have a history of epilepsy or seizures, current or past history of schizophrenia, metal implants or shrapnel in your head, or history of previous adverse events with TMS. If you are a female, you should not participate if you are pregnant or plan on becoming pregnant during your participation in this experiment. You must be using an effective form of birth control (e.g. birth control pills, surgically sterilized, IUD, cervical cap with a spermicide, or abstinence), and you must be willing to take a pregnancy test before being accepted into the research study. You must be living with HIV/AIDS to be in the study.

# WHERE WILL THE STUDY TAKE PLACE AND WHAT IS THE TOTAL AMOUNT OF TIME INVOLVED?

Firstly, a brain scan will be scheduled at the Magnetic Resonance Imaging and Spectroscopy Center (MRISC) situated on 740 Rose Street, Lexington 40536. This brain scan session will last an hour. All other research procedures will be conducted at the TMS Research Suite, Department of Psychiatry, 245 Fountain Court, Lexington, Kentucky 40509. You will need to come in once for the study. This visit will take 3 hours and then we will transport you to MRISC for another brain scan session after the TMS session at 245 Fountain Court. This scan session will also last one hour. The total amount of time you will be asked to volunteer for this study is 10-12 hours over the course of three days.

## WHAT WILL YOU BE ASKED TO DO?

If you agree to take part in this study, in your first visit, you will be asked to sign and date this consent form prior to any procedures. The table below highlights which days study activities will take place and whether they happen before or after the TMS session. If you are a woman of childbearing potential, you will also undergo a urine test to make sure you are not pregnant. Then we will ask you to get a brain MRI scan on day one. MRI uses magnetic fields to measure brain structure and brain activity. It involves lying down on a padded platform that is loaded into the circular center of the MRI machine. During a scanning session, you will be asked to remain still as images of your brain are acquired. You will be instructed to remove all jewelry and other metal-containing objects. Because the magnetic field will affect any metallic object, you should not participate if you have any type of metallic implant in your body, including pacemakers, aneurysm clips, shrapnel, metal fragments, orthopedic pins, screws, or plates, IUD's, or piercings that you cannot remove. On days two and three, we will assess your craving to smoke cigarettes. We will administer scales to assess craving and impulsive behavior.

| Study Task | Study Day | Before TMS | After TMS |
|----------------------------|-----------|------------|-----------|
| Pregnancy Test | 1 | Yes | No |
| MRI brain at MRISC | 1,2,3 | Yes | Yes |
| Motor Threshold | 1 | Yes | No |
| Cognitive tasks (computer) | 2,3 | Yes | Yes |
| Craving questionnaire | 2,3 | Yes | Yes |

On days two and three of the study will be the TMS sessions. You will receive both actual TMS and sham TMS in this study, on separate days. There are two groups in

this study. One group will receive the actual TMS first and the sham TMS later. The other group will receive sham TMS first and active TMS later. The TMS paradigm we will use is called theta burst stimulation (TBS) which is a short, and efficient TMS stimulation method. In the placebo group, you will receive a different kind of stimulation which mimics the actual experimental one but does not deliver any electricity to the brain. Before the TMS sessions, we will have you perform a few computer cognitive tests, craving and impulsivity scales.

The TMS equipment consists of an electric stimulator and a wire coil. Turning the stimulator on and off produces brief electrical currents in the coil, and these currents create a short-lived magnetic field around that coil (also called a 'magnetic pulse'). The wire coil is coated in plastic in order insulate the stimulator current, it is shaped like an '8', and it is a little larger than a letter-size piece of paper. When the coil is held close to the head, and it generates a magnetic pulse, the pulse can induce very small electric currents in the part of the brain that is closest to the coil. These currents are similar to the currents that the neurons in the brain produce when communicating with each other. By inducing these currents with the TMS coil, we can temporarily change the way that brain region functions, either making the region work harder or less hard. In this study, TMS will be used in a manner which is an investigational procedure, aimed at temporarily changing the way that a part of your brain works. TMS has been approved by the Food and Drug Administration (FDA) as a treatment for depression but in this study TMS is being

used to investigate if changes in the activities of certain areas of the brain affect memory. Although the form of TMS we use has not been approved by FDA for smoking cessation, another type of TMS called deep TMS has been approved by the FDA.

Before applying TMS, the study doctors will need to determine what strength of stimulation to use for you by establishing your personal "motor threshold" – a measure of the excitability of the area of the human brain called the motor cortex. To establish this threshold, the study doctor or a member of the study staff will first place the stimulator over the part of your brain that controls the motor activity in your right hand. You will hear a clicking sound and feel a tapping sensation at your scalp. The stimulator will be adjusted to give just enough energy so that the motor region of the brain sends signals to your hand muscles, to make your hand twitch. The smallest amount of energy required to make your hand twitch is called the "motor threshold." Everyone has a different motor threshold. This procedure will take about 20 minutes and will be done only on day one of the study. Then we will administer cognitive tests to assess how your brain makes decisions and chooses hypothetical rewards. You will also perform a visual attention test to assess how your eyes focus attention when seeing images related to smoking versus neutral images. You will then receive actual TMS versus placebo TMS depending on the group you were assigned to by chance initially. Both groups will get stimulation for 10 minutes.

For both active and sham TMS sessions, you will be seated comfortably in a chair, facing a computer screen placed about 5 feet away. Earplugs will be worn to protect your hearing. Your head will be held steady by a frame with a chin rest and the TMS coil holder frame, and study staff will ensure your comfort during the entire procedure. The study staff will administer the magnetic stimulation. You will be required to sit still while you receive the stimulation. To block out the clicking noise of the TMS procedure, we will provide you with earplugs. After the TMS session, you will then be administered the cognitive tests, craving and impulsivity scales again. Following this, we will transport you to MRISC for one more brain MRI scan.

## WHAT ARE THE POSSIBLE RISKS AND DISCOMFORTS?

Because of your participation in this study, you are at risk for the following side effects. You should discuss these with the researchers and your regular health care provider. The most serious known risk of TMS is the production of a convulsion (seizure). TMS procedures are associated with a very low risk of seizures. Out of tens of thousands of people given various forms of TMS to date, 16 people have been reported to have had a seizure. TMS can produce a convulsion when a series of pulses is given at high power and when repeated series of pulses are given extremely close together. This study will use only levels of TMS that are within safety guidelines. Levels of TMS that fall within the safety guidelines have not been associated with seizure in appropriately screened individuals. No seizures have occurred in normal volunteers with the dosage of TMS used in this study. To minimize this risk, we will medically screen you for any of the known characteristics that could lead to seizure. For example, if you have epilepsy you cannot participate in this study. You will be visually monitored during the TMS for any signs of seizure or muscle twitching. In spite of these precautions, there is a chance that you will experience a convulsion. Should this occur, our study doctor will be called and will assess if you need to be taken to the Emergency Department at UK Medical Center.

If you have a convulsion, you may require hospital admission and follow-up neurological evaluation. Having had a convulsion may make it difficult for you to obtain medical insurance, future employment, and to drive. It is not known whether having had one convulsion will make a person more prone to have future convulsions. Should you have a seizure caused by TMS in this protocol, we will provide you with a letter documenting that the seizure was experimentally induced.

The most common side effect of TMS is a "muscle-tension" type headache. We expect that about three out of ten people may experience a headache with the types of TMS used in this study. We will make every effort to reduce any discomfort by adjusting the position of the TMS coil on your head, altering the stimulation output of the coil, or taking breaks as required. If a headache occurs, it usually starts during or immediately after the TMS and lasts from minutes to hours after TMS. The headache usually goes away with standard over-the-counter pain medications. Neck pain may also occur. You may also experience some discomfort on your head where the coil is held. This is due to contraction of scalp muscles. Temporary numbness of the face has also been reported in rare instances that may last for several weeks after treatment.

The click noises produced by the TMS procedure are loud enough to be damaging to your ears. You will therefore be required to wear earplugs, provided by the experimenter. Additional side effects considered to be rare in TMS are dizziness, memory impairment, trouble concentrating, and acute mood changes. If these occur, these effects

do not last long (minutes to hours, but not day) and will resolve without need for treatment. There may be other risks that are currently unknown. The long-term effects of TMS are not known. There is also a risk of potential loss of confidentiality. Every effort will be made to keep your information confidential; however, this cannot be guaranteed.

While in the MRI scanner you may become too hot or too cold, in which case you may ask for an adjustment of room temperature or a blanket. Some people may become nervous or feel claustrophobic while in the scanner. If this happens, you may ask to be withdrawn and will be removed from the scanner immediately. A small number of people experience a sense of dizziness or vertigo while in the scanner due to the magnetic field. If this occurs and disturbs you, you may ask to be withdrawn and you will be removed immediately.

There is always a chance that any research procedure can harm you. The research procedures in this study are no different. In addition to risks described in this consent, you may experience a previously unknown risk or side effect. If you experience any adverse events (a bad effect) after leaving the study, please contact Gopalkumar Rakesh MD, Assistant Professor, Department of Psychiatry at 857-222-2276 during regular business hours. If outside regular business hours, please contact the Psychiatry department On Call Group at (859) 226-7063 and explain to the physician that you are a study participant. For women of child-bearing potential: The risks of exposure to magnetic fields during pregnancy are unknown. Women of childbearing capacity will be asked to take a pregnancy test before exposure to MRI. You will be excluded from the study if the test indicates that you may be pregnant.

# WILL YOU BENEFIT FROM TAKING PART IN THIS STUDY?

You may benefit from taking part in this study in helping you stop smoking. The study will inform us about how transcranial magnetic stimulation affects cognitive functions, visual attention, craving and impulsivity in people living with HIV.

## IF YOU DON'T WANT TO TAKE PART IN THE STUDY, ARE THERE OTHER CHOICES?

If you do not want to be in the study, there are no other choices except not to take part in the study.

## WHAT WILL IT COST YOU TO PARTICIPATE?

The University of Kentucky will not bill your insurance company, Medicare, or Medicaid for the study as it is done strictly for research. You will not incur any costs, should you decide to participate in this study.

# WHO WILL SEE THE INFORMATION THAT YOU GIVE?

Every effort will be made to maintain the confidentiality of your study records. We will make every effort to prevent anyone who is not on the research staff from knowing that you gave us information, or what that information is. When we write about or share the results from the study, we will write about the combined information. We will keep your name and other identifying information private. All your personal details will be stored separate from all other research data in an encrypted format. Your identity will remain confidential, unless you give prior written approval or unless it is required by law. Your name, address and social security number will be listed on the receipt for payment that you receive, as required by the Internal Revenue Service (IRS); but no information about your participation in this research project will be released. The study will also be registered on www.clinicaltrials.gov and collective data on number of patients recruited into this trial will be reported on the website. To ensure the study is conducted properly, officials of University of Kentucky may look at or copy pertinent portions of records that identify you.

You should know that in some cases we may have to show your information to other people because

For example, the law may require us to share your information with:

- a court or agencies, if you have a reportable disease/condition;
- Authorities, if you report information about a child being abused; or if you pose a danger to yourself or someone else.

To help us protect your privacy, this research has a Certificate of Confidentiality. The researchers can use this Certificate to refuse to disclose information that may identify you to anyone not connected with this study, or in any legal proceedings. The exceptions to this rule are release of information:

• you have requested us to provide, for instance, to your insurance company or doctor;

- to the sponsor (e.g., National Institutes of Health) or agency auditing the research (e.g., Food and Drug Administration);
- about child or elder abuse, neglect, or harm to yourself or others; and
- about you if it involves a reportable disease.

This policy does not prevent you from releasing information about your own participation in this study.

## CAN YOU CHOOSE TO WITHDRAW FROM THE STUDY EARLY?

You can choose to leave the study at any time. You will not be treated differently if you decide to stop taking part in the study. If you decide to withdraw from the study early, you will not receive any of the completion allowance described below. The data collected until that point of withdrawal from the study will remain in the study database and may not be removed. The study investigators can discontinue your participation for the following reasons: (1) if you verbally or physically assault another volunteer, patient or staff member at 245 Fountain Court; (2) if your behavior is disruptive to the other volunteers, patients, research staff or medical staff at 245 Fountain Court; (3) failure to comply with the alcohol, and drug use restrictions; (4) failure to comply with the pregnancy restrictions; (5) failure to complete a scheduled experimental sessions; (6) failure to perform the behavioral tasks to the best of your ability. If you are discharged from the study for any of these reasons, you will not receive the completion allowance described below. The medical doctor on this project can terminate your participation if he/she does not feel that it is medically safe for you to continue. If you experience intractable headaches with TMS, you can withdraw from the study with no ramifications to your clinic appointments. If your participation is terminated for medical reasons, you will receive the completion allowance for each of the sessions you completed.

# ARE YOU PARTICIPATING, OR CAN YOU PARTICIPATE, IN ANOTHER RESEARCH STUDY AT THE SAME TIME AS PARTICIPATING IN THIS ONE?

You may take part in this study if you are currently involved in another research study. It is important to let the investigator/your doctor know if you are in another research study. You should discuss this with the investigator/your doctor before you agree to participate in another research study while you are in this study.

## WHAT HAPPENS IF YOU GET HURT OR SICK DURING THE STUDY?

If you believe you are hurt or get sick because of something that is done in this study, you should immediately call Gopalkumar Rakesh MD, Assistant Professor, Department of Psychiatry at 857-222-2276. After business hours, please call the Psychiatry department On Call Group at (859) 226-7063 and explain to the physician that you are a study participant. The physician will determine what type of treatment, if any, is best for you at that time.

It is important for you to understand that the University of Kentucky does not have funds set aside to pay for the cost of any care or treatment that might be necessary because you get hurt or sick while taking part in this study. Also, the University of Kentucky will not pay for any wages you may lose if you are harmed by this study.

Medical costs related to your care and treatment because of study-related harm will be your responsibility. You do not give up your legal rights by signing this form.

#### WILL YOU RECEIVE ANY REWARDS FOR TAKING PART IN THIS STUDY?

For the first two days of the study, you will receive \$120 and for participation in the third day of the study, you will receive \$150.

With a few exceptions, study payments are considered taxable income reportable to the Internal Review Service (IRS). A form 1099 will be sent to you if your total payments for research participation are \$600 or more in a calendar year.

# WHAT IF NEW INFORMATION IS LEARNED DURING THE STUDY THAT MIGHT AFFECT YOUR DECISION TO PARTICIPATE?

We will tell you if we learn new information that could change your mind about staying in the study. We may ask you to sign a new consent form if the information is provided to you after you have joined the study.

## WILL YOU BE GIVEN INDIVIDUAL RESULTS FROM THE RESEARCH TESTS?

The investigators on this project will share with you any significant new findings that may develop during the course of your participation. At that time, you will be allowed to decide if you wish to continue in the study. If you choose not to continue, you will receive the completion allowance for each of the visits you attended.

## WILL WE CONTACT YOU WITH INFORMATION ABOUT PARTICIPATING IN FUTURE STUDIES?

The research staff would like to contact you in the future with information about participating in additional studies. If so, it will be limited to two times per year.

| | · | to be contacted in the future regarding your willingness to participate in future |
|---|---|---|
| research stud <b>Ves</b> | _ | Initials |

## WHAT ELSE DO YOU NEED TO KNOW?

Before you decide whether to accept this invitation to take part in this research study, please ask any questions now. Later, if you have questions about the study, you can contact the investigators directly at the phone numbers listed above. If you have concerns or questions about your rights and/or welfare as a volunteer in this research, you can contact the staff in the Office of Research Integrity at The University of Kentucky at (859) 257-9428 or toll free at 1-866-400-9428. We will give you a signed copy of this consent form to take with you.

A description of the clinical trial will be available on ClinicalTrials.gov as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# WILL YOUR INFORMATION (OR SPECIMEN SAMPLES) BE USED FOR FUTURE RESEARCH?

All identifiable information (e.g., your name, medical record number, or date of birth) will be removed from the information or samples collected in this study. This means that no link or code to your identity will be kept. After all identifiers have been removed, the information or samples may be used for future research or shared with other researchers without your additional informed consent, Once you give your permission to have your deidentified information or samples stored, they will be available indefinitely and cannot be removed due to the inability to identify them.

## **AUTHORIZATION TO USE OR DISCLOSE YOUR IDENTIFIABLE HEALTH INFORMATION**

The privacy law, HIPAA (Health Insurance Portability and Accountability Act), requires researchers to protect your health information. The following sections of the form describe how researchers may use your health information.

# Your health information that may be accessed, used and/or released includes:

Age, diagnoses of seizure disorder and schizophrenia if any, history of traumatic brain injury/loss of consciousness, medication history, duration of treatment with suboxone. The diagnoses in your chart will be looked at since these form part of inclusion criteria for the study. We would like to know how long you have been on suboxone as that would be used as a predictor variable in analyses of results from the study.

## The Researchers may use and share your health information with:

- The University of Kentucky's Institutional Review Board/Office of Research Integrity;
- Law enforcement agencies when required by law;
- University of Kentucky representatives;
- UK Hospital
- Food and Drug Administration

The researchers agree to only share your health information with the people listed in this document. Should your health information be released to anyone that is not regulated by the privacy law, your health information may be shared with others without your permission; however, the use of your health information may still be regulated by applicable federal and state laws.

You may not be allowed to participate in the research study if you do not sign this form. If you decide not to sign this form, it will not affect your:

Current or future healthcare at the University of Kentucky;

Page **6** of **8** 

- Current or future payments to the University of Kentucky;
- Ability to enroll in any health plans (if applicable); or
- Eligibility for benefits (if applicable).

After signing the form, you can change your mind and NOT let the researcher(s) collect or release your health information (revoke the Authorization). If you revoke the authorization:

- Send a written letter to: Gopalkumar Rakesh MD, Assistant Professor, Department of psychiatry, 2nd floor, 245 Fountain Court, Lexington 40509 to inform him of your decision.
- Researchers may use and release your health information already collected for this research study.
- Your protected health information may still be used and released should you have a bad reaction (adverse event).
- You will not be allowed to review the information collected for this research study until after the study is completed. When the study is over, you may have the right to access the information.

The use and sharing of your information has no time limit.

If you have not already received a copy of the Privacy Notice, you may request one. If you have any questions about your privacy rights, you should contact the University of Kentucky's Privacy Officer between the business hours of 8am and 5pm EST, Monday-Friday at (859) 323-1184.

# **INFORMED CONSENT SIGNATURES**

This consent includes the following:

- Key Information Page
- Detailed Consent

You will receive a copy of this consent form after it has been signed.

| Signature of research subject | Date |
|-------------------------------------------------------------|----------|
| Printed name of research subject | |
| Printed name of [authorized] person obtaining informed cons | sent and |

Attentional Bias Analyses. Attentional bias for cigarette cues will be calculated separately for each set of trials, by subtracting the average fixation time on neutral cues from the average fixation time on cigarette cues. Fixation time on cigarette cues for each session and resultant cigarette cue attentional bias score will be entered into separate linear fixed effects regression models. Dependent variables for these models will be fixation time on cigarette cues and attentional bias for cigarette cues respectively.

Cigarette craving analyses. TCQ-SF scores will be entered into a linear fixed effects regression model. Outcome variables for this model will be TCQ-SF score.

Resting state functional connectivity (rsFC) analyses. CONN functional connectivity toolbox (version 21.a) will be used for all preprocessing and neuroimaging analyses using standard procedures. Firstly, general linear model (GLM) analyses will explore if rsFC changed from two seeds (L. dlPFC and right insula) to all voxels following iTBS versus sham iTBS relative to baseline rsFC in participants who receive iTBS and sham iTBS. In first level analyses, a seed map will be created for every subject using respective seeds (L. dlPFC or right insula). In second level analyses, a between conditions contrast will be used to assess rsFC within-subject differences baseline, and following iTBS and sham ITBS. All second level analyses will use cluster level inferences based on Gaussian Random Field Theory. This will be done using general linear models (GLM) to generate a statistical map of t-values, that will subsequently threshold to reveal non overlapping clusters (<a href="https://web.conn-">https://web.conn-</a>

toolbox.org/fmri-methods/cluster-level-inferences). Two-sided p-values will be generated using cluster-level false discovery rate (FDR) correction <sup>62</sup>.